## TITLE:

Phase 2 study of OBP-301 (Telomelysin <sup>TM</sup>) in combination with Pembrolizumab and stereotactic body irradiation in patients with head and neck squamous cell carcinoma with inoperable, recurrent or progressive disease

**IRB Protocol #:** 19-12021148

IND #: 26377

**Version 3, Date:** 5/7/21

**Principal Investigators:** Doru Paul, MD, PhD

Weill Cornell Medical Center 1305 York Avenue, 12<sup>th</sup> Floor

New York, NY 10021 Phone 646-962-6200 Fax 646-962-1607

dop9054@med.cornell.edu

Statistician:

Paul Christos, PhD, Healthcare Pol & Res Director of the Research Design and

Biostatistics Core 402 E 67<sup>th</sup> St, Rm 234

646-962-8018

pac2001@med.cornell.edu

**Participating Sites:** *List all participating sites (include site name, PI, and contact information).* 

| Principal Investigator(s) | Academic Center(s) |
|---------------------------|-------------------------------|
| Doru Paul | Weill Cornell Medical College |
| Maged Ghaly | Northwell Health |
| Doug Adkins | Washington University |

## **Confidentiality Statement**

This document is confidential and is to be distributed for review only to investigators, potential investigators, consultants, study staff, Investigational Product supplier (Oncolys BioPharma Inc.)

## Page 3 of 99

Joint Clinical Trials Office (JCTO)

and applicable independent ethics committees or institutional review boards. The contents of this document shall not be disclosed to others without written authorization from WCM.

## **TABLE OF CONTENTS**

| 1 | STUDY SYNOPSIS | 13 | , |
|---|----------------|----|---|
| 2 | CTUDY CCHEMA | 21 | |

| 3 | F | BACKGROUND | 22 |
|---|---|---|---|
| 1.1 | The rati | onale for using a triple therapy combination in head and neck cancer | 22 |
| 1.4. | 1 Non-C | Clinical Studies | 30 |
| | 1.4.2 ( | Clinical Studies | 32 |
| 3.5 | Su | mmary of Potential Risks and Benefits | 35 |
| 3.6 | Do | osage and Treatment Periods | 36 |
| 3.7 | Pa | tient Population | 36 |
| 4 | ( | OBJECTIVES | 37 |
| 5 | S | STUDY DESIGN | 37 |
| 5.1 | Str | ıdy Overview | 37 |
| 6 | S | STUDY POPULATION | 39 |
| 6.1 | Se | lection of Study Population | 39 |
| 6.2 | Inc | clusion Criteria | 39 |
| 6.3 | Ex | clusion criteria | 41 |
| | 6.3 | 3.1 Patient Registration – Part 1 (WCMC Only) | 42 |
| | 6.3 | 3.2 Patient Registration – Part 2 (All Sites) | 42 |
| 6.4 | Sto | opping Criteria | 42 |
| | 6.4.1 | Patient Withdrawal Criteria | 42 |
| | 6.4.2 | Termination or Suspension of the Study | 43 |
| 7 | S | STUDY TREATMENTS | 44 |
| 7.1 | Inv | vestigational Product (IP) Identification | 44 |
| 7.2 | Do | osage and Treatment | 44 |
| 7.3 | Inv | vestigational product | 45 |
| | 5.3.1 S | tudy Supplies OBP-301 | 45 |
| | 7.3.2 | Selection and Timing and IT Administration for each Patient | 47 |
| | 7.3.3 | Injection Procedures | 48 |
| 7.4 | Pe | mbrolizumab | 51 |
| | 7.4.1 | General Concomitant Medication and Supportive Care Guidelines | 53 |
| | 7.4.2 | Rescue Medications & Supportive Care | 54 |
| 7.5 | Ra | diation therapy | 58 |
| 8 | S | TUDY PROCEDURES | 62 |
| 8.1 | Sc | hedule of Events | 63 |
| | 8.1.1 | Screening Visit | 65 |
| | 812 | Treatment Phase | 65 |

| | 8.1.3 | Follow up Phase | 65 |
|---|---|---|---|
| | 8.1.4 | Patient Withdrawal Criteria | 65 |
| 8.2 | In | Formed Consent Form (see appendix) | 67 |
| 8.3 | De | emographic Data and Baseline Characteristics | 67 |
| 8.4 | M | edical History, Concomitant Disease, Previous and Ongoing Medications | 67 |
| 8.5 | Sa | fety Assessments | 68 |
| | 8.5.1 | Adverse Events | 68 |
| | 8.5.2 | Physical Examination | 68 |
| | 8.5.3 | Vital Signs | 68 |
| | 8.5.4 | Electrocardiogram | 68 |
| | 8.5.5 | Laboratory Assessments | 69 |
| 8.6 | Ef | ficacy Assessments | 70 |
| | 8.6.1 | Imaging Assessment for the Study | 70 |
| | 8.6.2 | Definitions of Measurable and Non-Measurable Disease | 70 |
| | 8.6.3 | Response Criteria | 70 |
| | 8.6.4 | Determination of Tumor Stage According to Tumor, Lymph Nodes, Metasta (TNM) Classification | |
| 8.7 | Bi | opsies and Immune Monitoring (optional) | 72 |
| 9 | A | ADVERSE EVENTS | 72 |
| 9.1 | De | finitions | 72 |
| | 9.1.1 | Definition of an Adverse Event | 72 |
| | 9.1.2 | Severity of an Adverse Event | 73 |
| | 9.1.3 | Causal Relationship of an Adverse Event | 73 |
| | 9.1.4 | Definition of a Serious Adverse Event | 74 |
| | 9.1.5 | Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events and Serious Adverse Events | 75 |
| 9.2 | Do | ocumenting Adverse Events | 75 |
| | 9.2.1 | Recording of Adverse Events | 76 |
| | 9.2.2 | Reporting of AE to WCMC IRB | 76 |
| | 9.2.3 | Follow-up of Adverse Events and Serious Adverse Events | 76 |
| | 9.2.4 | Reporting of SAE to IRB | 76 |
| | d. For | multicenter studies, the multicenter core within the Quality Assurance Unit (QAU) will distribute the IND Safety Report | 77 |
| | 9.2.5 | Notification of Serious Adverse Event to Oncolys | 77 |
| | 9.2.6 | Notification of Suspected Unexpected Adverse Reactions | 78 |

| | 9.2.7 | Notification of Pregnancies | 78 |
|---|---|---|---|
| 9.3 | Μι | llticenter Study Monitoring | 78 |
| 10 | S | TATISTICAL ANALYSES | 78 |
| 10.1 | Ge | neral Considerations | 78 |
| 10.2 | De | finitions for Statistical Data Analysis | 79 |
| 10.3 | На | ndling of Missing Values and of Values outside the Detection Limits | 79 |
| | 10.3.1 | Data Collection | 79 |
| | 10.3.2 | REDCap | 79 |
| 10.4 | An | alysis Populations | 79 |
| | 10.4.1 | Safety Population | 79 |
| | 10.4.2 | Evaluable Population | 80 |
| | 10.4.3 | Intent-to-Treat (ITT) Population | 80 |
| | 10.4.4 | Per-Protocol (PP) Population | 80 |
| 10.5 | Eff | icacy Analysis | 80 |
| | 10.5.1 | Primary Efficacy Endpoint | 80 |
| | 10.5.2 | Secondary Efficacy Endpoints | 80 |
| | 10.5.3 | Exploratory Analysis | 81 |
| 10.6 | Co | rrelative Studies | 81 |
| 10.7 | Sat | ety Analyses | 84 |
| | 10.7.1 | Safety Endpoints | 84 |
| | 10.7.2 | Summary of Adverse Events | 84 |
| | 10.7.3 | Summary of Laboratory Assessments | 85 |
| | 10.7.4 | Summary of Special Laboratory Assessments | 85 |
| | 10.7.5 | Summary of Vital Signs | 85 |
| | 10.7.6 | Summary of Physical Examinations | 85 |
| | 10.7.7 | Summary of ECG Measurements | 85 |
| | 10.7.8 | Concomitant Medications | 85 |
| | 10.7.9 | Adverse Event Stopping Rule | 85 |
| 10.8 | De | termination of Sample Size | 87 |
| 11 | R | EGULATORY REQUIREMENTS | 89 |
| 11.1 | Re | gulatory Approvals | 89 |
| 11.2 | Ins | titutional Review Board/Ethics Committee Approval | 89 |
| 11.3 | Eth | nical Conduct of the Study | 89 |
| 11.4 | Pai | ticipant Informed Consent | 90 |

| 11.5 | Compliance with Trial Registration and Results Posting Requirements | 90 |
|---|---|---|
| 12 | Data and Safety Monitoring Plan (DSMP) | 91 |
| 13 | ADMINISTRATIVE PROCEDURES | 91 |
| 13.1 | Financing, Liability/Indemnity/Insurance | 91 |
| 13.2 | Recording of Data and Retention of Records | 91 |
| 13.3 | Retention of Records | 92 |
| 13.4 | Disclosure and Data Confidentiality | 92 |
| 13.5 | Publication of Results | 92 |
| 14 | CLINICAL STUDY REPORT | 92 |
| 15 | AppendixES | 93 |
| 15.1 | ECOG performance status | 93 |
| 15.2 | Comparison of RECIST 1.1 and iRECIST | 93 |
| 15.3 | Annendix | 94 |

## LIST OF ABBREVIATIONS

| Ad5 | adenovirus serotype 5 |
|-------|---------------------------------------------|
| AE | adverse event |
| AJCC | American Joint Commission on Cancer |
| ALT | alanine transaminase |
| APC | antigen presenting cell |
| AST | aspartate transaminase |
| BSLD | baseline sum longest diameters |
| CAR | Coxsackie adenovirus receptor |
| CBC | complete blood count |
| CBER | Center for Biologics Evaluation |
| cGMP | current Good Manufacturing Practice |
| CR | complete response |
| CRAd | Conditionally Replicative Adenovirus |
| CRF | case report form |
| eCRF | electronic case report form |
| CRO | contract research organization |
| CSR | clinical study report |
| СТ | computed tomography |
| CV | coefficient of variation |
| CTCAE | Common Toxicity Criteria for Adverse Events |
| DLT | dose-limiting toxicity |
| DNA | deoxyribonucleic acid |
| ECG | electrocardiogram |
| EDC | electronic data capture |

| FDA | Food and Drug Administration |
|--------|-----------------------------------------------------|
| FSH | follicle stimulating hormone |
| GCP | Good Clinical Practice |
| GEJ | Gastroesophageal Junction |
| GLP | Good Laboratory Practice |
| GM-CSF | granulocyte-macrophage colony stimulating factor |
| HBV | hepatitis B virus |
| HBsAg | hepatitis B surface antigen |
| HCV | hepatitis C virus |
| HED | human equivalent dose |
| НЕК | human embryonic kidney (cell) |
| HIPAA | Health Insurance Portability and Accountability Act |
| HIV | human immunodeficiency virus |
| hTERT | human telomerase reverse transcriptase |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| ICI | Immunotherapy with Checkpoint Inhibitors |
| IEC | independent ethics committee |
| IL | interleukin |
| IM | intramuscular |
| IMRT | Intensity-modulated Radiation Therapy |
| IND | Investigational New Drug |
| INR | international normalized ratio |
| IP | investigational product |
| irCR | immune-related complete response |

| irPD | immune related progressive disease |
|-------------------------|----------------------------------------------|
| irPR | immune-related partial response |
| irRC | immune-related response criteria |
| irSD | immune-related stable disease |
| IRB | institutional review board |
| IRES | internal ribosomal entry site |
| ITT | intent-to-treat |
| IV | intravenous |
| KPS | Karnofsky Performance Status Scale |
| LD | longest diameter |
| LDH | lactate dehydrogenase |
| LLOQ | lower limit of quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MFD | maximum feasible dose |
| MRI | magnetic resonance imaging |
| mRNA | messenger RNA |
| MTD | maximum tolerated dose |
| NCI | National Cancer Institute |
| NOAEL | no adverse effect level |
| NOEL | no effect level |
| NTL | non-target lesion |
| OBP-301 (Telomelysin ™) | OBP-301 |
| ORR | objective response rate |
| os | overall survival |
| PD | progressive disease |

| PD-L1 | Programmed death-ligand 1 |
|---|---|
| PFS | progression free survival |
| PI | Principal Investigator |
| PP | per-protocol |
| PR | partial response |
| PTT | prothrombin time |
| qPCR | quantitative polymerase chain reaction |
| RECIST | response evaluation criteria in solid tumors |
| iRECIST | Immune response evaluation criteria in solid tumors |
| RNA | ribonucleic acid |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SBRT | Stereotactic Body Radiation Therapy |
| SOP | standard operating procedure |
| SUSAR | suspected unexpected adverse reaction |
| TIL | tumor infiltrating lymphocytes |
| TL | target lesion |
| TNF | tumor necrosis factor |
| TNM | tumor; lymph nodes; metastasis: classification of malignant tumors |
| $T_{\rm reg}$ | regulatory T cell |
| TTR | time to treatment response |
| T-VEC | talimogene laherparepvec |
| US | United States |
| USP | United States Pharmacopoeia |

| ULN | upper limit of normal |
|------|-------------------------------|
| VP | viral particles |
| WCM | Weill Cornell Medicine |
| WCMC | Weill Cornell Medical College |
| XTT | cell viability assay |

## 1 STUDY SYNOPSIS

| Protocol Title: | Phase 2 study of OBP-301 (Telomelysin <sup>TM</sup> ) in combination with Pembrolizumab and stereotactic body irradiation in patients with head and neck squamous cell carcinoma with inoperable, recurrent or progressive disease. |
|---|---|
| Protocol Number: | |
| Study Sites: | <ol> <li>Weill Cornell Medical College</li> <li>Northwell Health</li> <li>Washington University</li> <li>4.</li> </ol> |
| Study Phase: | Phase II |
| Study | Primary Objective: |
| Objective(s): | To examine the ORR of OBP-301 in combination with<br>pembrolizumab and SBRT in advanced head and neck<br>squamous cell cancer as assessed by the RECIST 1.1<br>response rate. |
| | <ul> <li>To evaluate the safety of the combination of multiple<br/>intratumoral injections of OBP-301 with SBRT and<br/>pembrolizumab.</li> </ul> |
| | Secondary Objectives: |
| | To examine other measures of efficacy of the combination of OBP-301 intratumoral injections in combination with SBRT and pembrolizumab in recurrent, inoperable or progressive HNSCC including the disease control rate, duration of response, overall survival and progression free survival. |
| | Exploratory Objectives (optional): |
| | Patients undergoing treatment with OBP-301 will have standard fine needle tissue biopsies along with correlative blood samples. In order to observe a potential response in the non-injected lesions, if several tumors are present, biopsies will be taken both from an injected tumor and a non-injected tumor and a comparison will be done between them. |
| | <ul> <li>To determine viral related biomarkers in the tumor: i.e. proof of the presence of the replicating virus (i.e-Adenovirus Hexon Protein) in the tumoral tissue.</li> <li>To examine the tumor-immune microenvironment prior to and following OBP-301, SBRT and pembrolizumab therapy.</li> </ul> |

| • | To examine treatment response to OBP-301 + SBRT + |
|---|-------------------------------------------------------|
| | pembrolizumab by monitoring changes in plasma and |
| | tumor tissue-derived exosomes and circulating tumoral |
| | DNA. |

- To examine and characterize the intra-tumoral and systemic immune responses by multi-parameter flow cytometry.
- To determine changes in circulating tumor cells as quantified by the TelomeScan, a liquid Biopsy diagnostic tool. The blood of 10 patients at a maximum of 4 time points will be analyzed.

## **Study Design:**

This is a phase II study of OBP-301 in combination with pembrolizumab and SBRT (or equivalent) in advanced HNSCC which is either recurrent and inoperable, or progressing after prior radiation with curative-intent for advanced disease (adjuvant or definitive with or without chemotherapy or cetuximab).

The efficacy of pembrolizumab monotherapy is modest in second or third line of treatment of advanced head and neck cancer (~response rate 16-22%). SBRT reirradiation in patients that received prior surgery and chemoradiation for advanced disease is associated with a RR of approximately 60% and approximately 50% 1-year survival. Recently, the results of the Keynote-048 study were published. The projected 1-year survival in the immunotherapy arms with pembrolizumab alone or pembrolizumab and chemotherapy was approximately 57%. So, at present, the benchmark RR for patients with head and neck squamous cell carcinoma with inoperable, recurrent or progressive disease treated with SBRT is approximately 60% and the 1 year survival for patients with head and neck squamous cell carcinoma with inoperable, recurrent or progressive disease using the most effective contemporary treatments including immunotherapy is approximately 50-57%. Trying to improve the results of the current standard of care, this study will examine the effects of oncolytic virus, OBP-301, administered in addition to pembrolizumab and SBRT in this patient population.

A total of 36 patients will be enrolled into a two-stage parallel cohort design: In the first stage, 12 patients will be enrolled.

All patients will receive intratumoral injection(s) with OBP-301 in a level 2 biohazard room by an experienced ENT surgeon. If tolerated and no progression is observed, up to twelve injections may be given in each patient.

The volume of OBP-301/tumor will be dependent on the targeted tumor volume. The same concentration of OBP-301 will be used for all patients  $(1 \times 10^{12} \text{ yp/ml})$ .

A maximum volume of 4 ml or 4 x10<sup>12</sup> vp total OBP-301 dose per treatment day will be administered. This maximum volume will be divided among one or more injectable lesions with the largest lesion getting the largest dose portion. The OBP-301 dose distribution between tumors will be at the discretion of the Investigator. (please see detailed description Section 5.3.2 Table 1).

If the targeted injected lesion(s) disappear, another lesion can be injected at the Investigator's discretion.

## **Treatment schedule is as follows:**

- **D1:** Targeted tumor(s) will be injected with intratumoral OBP-301 alone.
- **D8:** Patients will receive both intratumoral OBP-301 and systemic pembrolizumab.
- **D15- D29**: Radiotherapy with SBRT (or equivalent) will be given for a total of 5 doses on days 15, 18, 22, 25, 29
- **D15-D29:** Concurrent with radiation intratumoral OBP-301 injections to targeted tumor(s) will be given on days 18 and 25

## There will be no concurrent pembrolizumab given during SBRT.

D31: Systemic pembrolizumab will be resumed on a standard every 21-day schedule with concurrent intratumoral injections of OBP-301 on the same treatment day.

A minimum additional 3 doses of concurrent OBP-301 and pembrolizumab will be given [day 73] if no toxicity, technical impediment to injection or progression is seen.

A maximum total of up to 9 doses of concurrent OBP-301 and pembrolizumab will be given [day 183].

Pembrolizumab alone will be continued after day 183 for a total treatment time up to 1 year.

# Investigational Product Administration:

OBP-301, the investigational product (IP) is formulated in 20 mM Tris pH 8.0, 25 mM NaCl with 2.5% glycerin, USP by volume. OBP-301 will be injected into the target tumor lesions.

OBP-301  $(1 \times 10^{12} \text{ VP/mL})$  will be administered as intratumoral injection cutaneous, subcutaneous, and nodal tumoral lesions that are deemed safe for percutaneous or transmucosal injection therapy by the study Investigators.

At least one measurable lesion will be designated as a targeted lesion for intratumoral injection with OBP-301 and will be monitored for response. ORR will take into consideration all lesions injected or not.

| Planned Patients: | A maximum of 36 eligible patients will be enrolled in the study. |
|---|---|
| Participant Selection Criteria: | <ul> <li>Inclusion Criteria:</li> <li>Patients who meet all of the following criteria will be considered for inclusion in the study: <ol> <li>Be willing and able to provide written informed consent/assent for the trial.</li> <li>Be ≥18 years of age on the day of signing the informed consent.</li> <li>Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.</li> <li>Have histologically or cytologically confirmed advanced head and neck squamous cell cancer with cutaneous, subcutaneous or nodal tumors deemed as injectable lesions [see definition below] and have measurable disease for the primary study endpoint of overall response rate by RECIST 1.1 and iRECIST. In addition they must have: <ol> <li>A.1. A single measurable tumor at least 1 cm in size and amenable to intratumoral injection or</li> <li>Multiple measurable tumors that in aggregate have a longest diameter of ≥ 10 mm</li> </ol> </li> </ol></li></ul> |
| | <ul> <li>Note: Injectable lesion definitions: lesions amenable to percutaneous approach, if technically feasible</li> <li>5. Recurrent and inoperable tumor, progressing after prior radiation with curative-intent for advanced disease (adjuvant or definitive with or without chemotherapy or cetuximab). No prior treatment for local regional recurrence (LRR).</li> <li>6. Tumors may be either HPV+ or HPV</li> <li>7. Tumor must be PD-L1 positive, defined as CPS ≥ 1.</li> <li>8. Be willing to provide tissue; newly obtained biopsy specimens or formalin-fixed, paraffin-embedded (FFPE) block specimens.</li> <li>9. Female subjects of childbearing potential have a negative urine or serum pregnancy test within 14 days prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. It is permissible for this serum test to be performed on the same day, within 14 days prior to enrollment. And male / female subjects of childbearing potential must agree to use an adequate method of contraception starting with signing the informed consent through 120 days after the last dose of study medication.</li> <li>10. Demonstrated adequate organ function as defined in following criteria. All screening labs should be</li> </ul> |

performed within 14 days of enrollment. Note: Subject must not have taken transfusion, hematopoietic agent; granulocyte-colony stimulating factor (G-CSF) etc., and/or oxygen supplementation within 7 days before the screening labs.

- A) Absolute neutrophil count (ANC)>=1,000 /mm3
- B) Platelets>=100,000 /mm3
- C) Hemoglobin>=9.0 g/dL
- D) Serum total bilirubin<=2.0 mg/dL
- E) Aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT) (SGPT) <= 2.5x Upper limit of normal (ULN). For subjects with liver metastases<= 5x ULN.
- F) Serum creatinine<= 1.5 mg/dL; or if serum creatinine >1.5 mg/dL, measured or calculated creatinine/clearance>=60 mL/min (Cockcroft-Gault formula).
- 11. Life expectancy of  $\geq 6$  months from the first OBP-301 treatment.
- 12. Understand the study requirements and the treatment procedures, and is willing to comply with all specified follow- up evaluations, and provides written informed consent before any study-specific tests or procedures are performed.

#### **Exclusion Criteria:**

The presence of any of the following criteria will constitute cause for the exclusion of the participant:

- 1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 2 weeks (chemotherapy, small molecule), or 3 weeks (antibody) of study Day 1.
- 2. Has an active autoimmune disease that has required systemic treatment in past 2 years.
- 3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (greater than the equivalent of prednisone 20 mg/day) or any other form of immunosuppressive therapy within 7 days prior to study Day 1. Daily dose of maintenance prednisone 10mg or equivalent is allowable.
- 4. Has a known additional malignancy that is progressing or requires active treatment, with the exception of stable/low grade tumors that are not expected to influence life-expectancy (e.g. skin SCC, basal cell, differentiated thyroid cancer, prostate cancer on hormonal therapy).
- 5. Has received a live vaccine within 30 days of planned start of study therapy.

- 6. Has a known history of Human Immunodeficiency Virus.
- 7. Has known active Hepatitis B or Hepatitis C.
- 8. Has known history of, or any evidence of active, non-infectious pneumonitis.
- 9. Has an active infection requiring systemic therapy.
- 10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
- 11. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
- 12. Previous severe hypersensitivity to another monoclonal antibody.
- 13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
- 14. Prior intolerance related to severe (>=grade 3) irAE to a prior anti-immune checkpoint inhibitor agent leading to discontinuation of anti-immune checkpoint inhibitor therapy.
- 15. Any disorder or condition, or any medication that would put the patient at risk from bleeding after direct tumor injection.
- 16. Not a candidate for SBRT (or equivalent) given for potentially curative intent. All tumors must receive SBRT. For example, patients with locoregional neck recurrence without significant overlap with the previous radiation field, and who do not warrant SBRT for reirradiation as per the treating radiation oncologist (e.g. out-of-field recurrence), will not be included in the study.
- 17. Received prior immunotherapy with checkpoint inhibitors or other immunotherapy agents.
- 18. Exclude injection of study agent adjacent to great vessels
- 19. Exclude injection into tumor impinging tracheostomy sites
- 20. Exclude subjects with history of bleeding diathesis
- 21. Exclude patients with abnormal coagulation profile (PT/PTT).
- 22. Exclude subjects that have been treated with two or more courses of radiation therapy to the head and neck, including patients who previously received palliative reirradiation for recurrence.

| Study Procedures: | <ol> <li>OBP-301 1.0-4.0x10<sup>12</sup> viral particle/treatment day delivered by intratumoral injection therapy into one or more tumors per study schedule.</li> <li>SBRT (or equivalent) 40-45 Gy divided over a total of 5 treatments.</li> <li>Pembrolizumab 200 mg intravenous per study schedule.</li> </ol> |
|---|---|
| Study Endpoints: | Primary Endpoint: |
| | • To examine the efficacy of OBP-301 in combination with pembrolizumab and SBRT in advanced head and neck squamous cell cancer as assessed by the RECIST 1.1 response rate |
| | To examine the safety of multiple OBP-301 intratumoral injections in combination with pembrolizumab or/and SBRT |
| | • Secondary Endpoints: |
| | To determine the following additional measures of efficacy including: |
| | Overall survival (OS) at 1 year |
| | <ul> <li>Progression free survival (PFS)</li> </ul> |
| | Disease control rate at 6 months |
| | Immune related Response Rate (irRR) |
| | Time to response in non-target lesions |
| | Exploratory Analysis (optional): |
| | Correlative endpoints include the following: |
| | <ul> <li>To examine the tumor-immune microenvironment prior to and following OBP-301, SBRT and pembrolizumab therapy both in injected and non-injected lesions.</li> <li>To examine treatment response to OBP-301 + SBRT + pembrolizumab by monitoring changes in plasma exosomes and circulating tumoral DNA.</li> </ul> |
| | <ul> <li>To examine and characterize the immune infiltrate by multi-parameter flow cytometry.</li> <li>To determine viral related biomarkers in the tumor: i.e.</li> </ul> |
| | proof of the presence of the replicating virus (i.e. |

Receptor (CAR).

tool.

Adenovirus Hexon Protein) in the tumoral tissue or/and presence of the receptor for Coxsackie Adenovirus

To determine changes in circulating tumor cells as quantified by the TelomeScan, a liquid Biopsy diagnostic

## Statistical Analysis:

The primary endpoint for this study will be the objective response rate (CR + PR). Sample size recommendations for the phase II design are determined according to Simon's two-stage design (Simon R, 1989). We project an objective response proportion of 61%, below which the response will be unacceptable, and an objective response proportion of 78%, above which the regimen will be considered worthy of further exploration. The null hypothesis that the objective response proportion is less than or equal to 61% will be tested against the alternative hypothesis that the response proportion is greater than or equal to 78%.

The sample size computations were performed assuming 10% level of significance and 80% power. In the first stage, 12 patients will enter the study. If 7 or fewer respond, the study will be terminated early and declared to have a negative result. If 8 or more patients respond, enrollment will be extended to 36 patients. At Stage 2, the treatment will be declared effective and worthy of further testing if 26 or more patients respond among the 36 patients entered. This two-stage design yields  $a \ge 0.80$  probability of a positive result if the true percentage of overall responders is  $\geq 78\%$ . It yields a  $\geq 0.90$ probability of a negative result if the true percentage of overall responders is  $\leq 61\%$ . A 95% confidence interval constructed around the expected objective response proportion of 78% can be estimated to be within  $\pm$  16.0% of the observed response proportion. Assuming 10% are unevaluable/ineligible, we anticipate that a total of 14 patients will be enrolled in the first stage, 40 in both the first and second stage if the study proceeds to the second stage.

**Statistical Table.** Numbers of observed responders required to accept or reject H0 at each stage. Under this design, H0 will not be rejected at Stage 1.

| | N | Accept H <sub>0</sub> | Reject H <sub>0</sub> |
|---------|----|-----------------------|-----------------------|
| Stage 1 | 12 | ≤ 7 | |
| Stage 2 | 36 | ≤25 | >26 |

## **Study Duration:**

Approximately 30 months

Screening evaluations may be conducted up to 4 weeks before the first anticipated OBP-301 administration. Each patient will be in the study for 30 months following the first intratumoral injection of OBP-301.

## 2 STUDY SCHEMA



#### 3 BACKGROUND

## 1.1 The rationale for using a triple therapy combination in head and neck cancer

The Programmed Death Ligand-1 (PD-L1) and its receptor (PD-1) are important regulators of T cell activity<sup>1</sup>, and their inhibitors have now demonstrated antitumor activity in several malignancies<sup>2,3</sup> including melanoma<sup>4,5</sup>, lung<sup>6-9</sup>, renal<sup>10</sup>, and bladder cancers<sup>11</sup>. Despite a high level of PD-L1 expression in head and neck tumors (up to 80%), progress in checkpoint inhibitors treatment of cancers of head and neck have been limited. The response rate of monotherapy with checkpoint inhibitors in second line recurrent or locally advanced head and neck cancers has been only13-18% across the different PD-1 inhibitors<sup>12-18,42</sup>.



FIGURE 1 Change from baseline of head and neck cancer tumors with pembrolizumab (Ref 13)

Although activity is relatively modest, some patients live longer and those that respond tend to have durable responses of 12 months or greater with few patients stopping therapy for an adverse event (**Fig 1**). In 2016 pembrolizumab and nivolumab have been approved for second line treatment of recurrent or locally advanced head and neck cancers

A novel concept in immuno-oncology is the use of cancer specific oncolytic viral therapy to induce an immunogenic cell death in the tumor to augment the immune activation driven by PD-1 inhibition. This involves selective replication within neoplastic cells, resulting in a direct lytic effect on tumor cells, and induction of systemic antitumor immunity  $^{19}$ . OBP-301 is a telomerase-specific, replication-selective adenovirus in which the human telomerase reverse transcriptase (hTERT) promoter drives viral replication efficiently killing only cancer cells  $^{20-23}$ . OBP-301 has been examined in a phase I study in solid tumor patients, with an established safe dose of  $1 \times 10^{12}$  viral particles/tumor injection. In this study, there was evidence of systemic immune response with the development of a neutralizing

antibody (Ab) response in all tested patients, and up regulation of serum IL-6 and IL-10 levels in 8/9 and 7/9 patients respectively<sup>24</sup>. Notably, 7/16 patients had stable disease at 56 days, suggesting preliminary efficacy. The most common side effects were local irritation and erythema from the injection (3/16 grade 3), as well as fever, chills, and fatigue (grade 1-2) in 30-40% of patients<sup>24</sup>.

There is preclinical and clinical evidence that OBP-502 (the murine version of OBP-301) is synergistic with anti-PD-1 therapy providing rationale for this proposal. (Figs 2A and 2B). In vitro and in vivo studies have shown the potential of OBP-502 to activate antitumor immunity, leading to sensitization of non-immunogenic gastrointestinal tumors to PD-1 antibody. The growth in vaccinated mice was significantly suppressed than control mice and there was induction of tumor-infiltrating cells following the administration of OBP-502 with an anti-PD1 antibody combination compared to pre injection. (Figures 2A and 2B and Ref 43).



Figure 2A Synergistic effects of OBP-502 and Anti-PD1 Antibody

■ In addition, a Japanese Phase I study of OBP-301 in combination with Anti-PD-1 is ongoing. (NCT03172819). The study aims to evaluate safety and potential efficacy of combination of OBP-301 and pembrolizumab in patients with advanced or metastatic solid tumors. Preliminary safety data in 9 evaluable patients demonstrated that the combination of OBP-301 and pembrolizumab was well tolerated in the tested dose of 1x10<sup>12</sup> vp/tumor. Most common adverse events included fever (grade 1-2) hepatic disorder (grade 1-3) and pleural effusion (grade 1). There were early signs of efficacy 3/9 partial response (PR)s<sup>44</sup>.



Figure 2B Induction of tumor-infiltrating cells was significantly increased following combination of OBP-502 and Anti-PD-1Ab.

Also, OBP-301 has a radiosensitizing effect. As shown **in Figure 3**, OBP-301 increases the effect of ionizing radiation in a dose dependent manner. OBP-301 sensitizes human cancer cells to ionizing radiation by inhibiting the radiation-induced DNA repair machinery, and also eliminates radio-resistant quiescent cancer stem-like cells by promoting cell cycle entry.



Figure 3 Radiosensitizing effect of OBP-301 and Anti-PD1 Antibody

An Investigator-initiated phase I/II Study of OBP-301 with radiation therapy in Japanese head and neck or/and thoracic malignant cancers patients unfit for surgery has been completed. Thirteen patients with esophageal cancer have been treated (3 at the highest dose level of 1X10<sup>12</sup>vp/tumor). Toxicities have been manageable. The only observed grade <sup>3</sup>/<sub>4</sub> toxicities have been leukopenia (8%) and lymphopenia (77%). Grade1/2 toxicities include transient fever without evidence of infection (62%), chills (15%), nausea (25%), esophagitis (31%), anorexia (39%) and pneumonitis (23%). Indication of reduction in area of treated tumor was observed in 11 (8 clinical CR and 3 PR) out of 12 evaluable patients (objective response rate: 91.7%). Pathological responses were also observed in 8 patients (66.7%)<sup>45</sup>.

Preclinical data in murine cancer models show improved tumor growth control and survival when radiation therapy (RT) is combined with a PD-1 inhibitor<sup>40</sup>.

Given the excellent toxicity profile of both checkpoint inhibitors and Radiation therapy and OBP-301 there is a rationale to combine OBP-301 with Radiation therapy and a checkpoint inhibitors.

## 1.2 Locally recurrent head and neck cancer (HNC)

Recurrent HNC in a previously irradiated field has a poor prognosis. When a recurrence develops in a head and neck cancer in an area previously treated with radiation, the mainstay of treatment remains local control of disease. The recurrence can have an attempt at salvage by surgery but this is often not possible given the extent of disease and previous therapy. A common approach involves re-irradiation to provide survival benefit over chemotherapy alone however the median survival in most series remains only 9-12 months with radiation only, depending upon patient and disease-related factors<sup>36</sup>. Treatment options are often limited. For unresectable disease, systemic therapy alone, the historical standard of care, results in 10–15% 1-year overall survival (OS) and virtually no long-term survivors<sup>36,37,38</sup>. In the EXTREME trial, only 3% (6/222) and 1% (2/220) of patients enrolled in the cetuximab and control arms, respectively, were known to still be alive after 5 years.<sup>38</sup>

For patients with recurrent or second primary HNC within a previously irradiated area, the only potentially curative option is a second course of radiation, with or without chemotherapy, termed reirradiation (RRT). Early experiences with RRT in selected patients demonstrated OS rates (30–50%) that compared favorably to chemotherapy alone<sup>39</sup>.

More recently, concomitant chemotherapy and stereotactic body irradiation (SBRT) has been adopted by some as a treatment strategy of choice for this patient population. Two consecutive multi-institutional cooperative group studies that used concurrent chemotherapy and re-irradiation for SCCHN, demonstrated the feasibility of re-irradiation. Two prospective studies<sup>32,33</sup> done by a French group have shown support for SBRT reirradiation. The first feasibility study<sup>32</sup> included 40 patients, with an SBRT dose of 36 Gy in 6 fractions, given over 11 to 12 days. The median OS was 13.6 months. There was a 79% response rate, and minimal toxicity (only G3 toxicity in 4 patients). Subsequently, the same group (Lartigau<sup>33</sup> et al.) published a multi-institutional phase II study of SBRT reirradiation (same dose/technique) with concurrent cetuximab in 56 patients and they found a response rate of 58.4%. The median OS was 11.8 months, the 1-year OS was 48%, and the median PFS was 7.1 months. Of 49 evaluable patients, 49% had a complete response and 20% had a partial response. Eighteen patients (32%) developed G3 or higher toxicity, and there was 1 death from hemorrhage. Two other retrospective studies<sup>34,35</sup> showed response rates ranging from 50% <sup>34</sup> to 80% <sup>35</sup> an OS at 1 year around 50% but higher severe late toxicity. A 2017 review of the most relevant SBRT studies showed that response rates to SBRT in the recurrent head and neck cancer setting are approximately  $60\%^{71}$ .

Recently, the Keynote-048 study was completed and the results were published<sup>67</sup>. The follow-up was only 11.5 months but the 1 projected year survival in the immunotherapy arms with pembrolizumab alone or pembrolizumab and chemotherapy was approximately 57%. So, the benchmark 1 year survival using the most effective treatments from the clinical studies completed so far is 50-57%.

At ASCO 2019, Harrington, K. J. et al. reported the safety and preliminary results of a Phase 1 B study<sup>46</sup> investigating the efficacy of another adenoviral construct, talimogene laherparepvec (T-VEC) administered locally in the tumor in combination with systemic pembrolizumab in patients with recurrent or metastatic squamous cell carcinoma of the head and neck. The primary objective was to evaluate safety, as assessed by the incidence of dose limiting toxicity (DLT). Key secondary objectives were objective response rate (ORR), best overall response per immune-related RECIST, and long-term safety. 36 pts were enrolled and treated: The ORR was 16.7% (6/36 pts; 5 PD-L1-positive; 95% CI, 6.4–32.8), and the disease control rate (objective response/stable disease) was 38.9% (14/36 pts; 11 PD-L1-positive; 95% CI, 23.1–56.5). The combination demonstrated a manageable safety profile. The same author suggested recently that radiotherapy approaches may add to this combination<sup>47</sup>.

## Unpublished experience:

A retrospective chart review of 20 patients treated in Northwell Health Monter Cancer Center with chemotherapy + SBRT or Cetuximab + SBRT confirmed the guarded prognosis of the majority of these patients.

In our cohort, median age of the patients was 71 years. 13 men and 7 women were treated with chemotherapy + SBRT or Cetuximab + SBRT. 5 patients received Cetuximab + SBRT and 15 patients received chemotherapy + SBRT. The maximum follow up time was 2 years.

- -35% (7/20) patients progressed very fast after the local ttx and lived an average of 3.5 months after the chemotherapy + SBRT or cetuximab + SBRT.
- -(50%) 10/20 patients were still alive but progressed after an average duration of 5.4 months.
- -15% (3/20) patients did not progress and were alive at a f/up of 7, 12, and respectively 14 months.

Similarly, the University of Chicago has shown in series of publication of re-irradiation (not SBRT, but hyper-fractionated radiation) of HNSCC that prognosis is guarded with only 15-20% of patients alive at 2 years (e.g. Seiwert et al JCO).

Clearly, there is an urgent need to improve the grim prognostic of patients with recurrent unresectable head and neck cancer that have been previously irradiated.

Conclusion and study rationale Treatment of recurrent unresectable head and neck cancer is an unmet medical need, for which drug development is lacking and for which currently

there is no standard of care. In the NCCN guidelines version 2.2018 it is clearly stated: "Research opportunities for reirradiation should be strongly considered in patients with unresectable head and neck cancer".

Given the proven radiosensitizing effects of OBP-301 and the synergistic interaction of OBP-301 with Pembrolizumab<sup>42</sup>, and the recent SBRT data in recurrent head and neck cancer<sup>46,47</sup> this is a clear opportunity for OBP-301 to be used together with SBRT and Pembrolizumab in the recurrent unresectable head and neck cancer setting. We believe that this triple local and systemic combined approach represents a powerful synergistic therapeutic modality to attack cancer both directly and, indirectly, by stimulating the immune system.

## 1.3 Oncolytic viral therapy background and rationale

A novel concept in immuno-oncology is the use of cancer specific oncolytic viral therapy to induce an immunogenic cell death in the tumor to augment the immune activation driven by PD1 inhibition. This involves selective replication within neoplastic cells, resulting in a direct lytic effect on tumor cells, and induction of systemic antitumor immunity<sup>19</sup>. OBP-301 is a telomerase specific, replication-selective adenovirus in which the human telomerase reverse transcriptase (hTERT) promoter drives viral replication efficiently killing only cancer cells <sup>20-23</sup>. OBP-301 has been examined in a phase I study in solid tumor patients, with an established safe dose of Ix10<sup>12</sup> viral particles/tumor injection. In this study, there was evidence of systemic immune response with the development of a neutralizing Ab response in all tested patients, and up regulation of serum IL-6 and IL-10 levels in 8/9 and 7/9 patient's respective<sup>24</sup>. Notably, 7/16 patients had stable disease at 56 days, suggesting preliminary efficacy. The most common side effects were local irritation and erythema from the injection (3/16 grade 3), as well as fever, chills, and fatigue (grade 1-2) in 30-40% of patients<sup>24</sup>. There is preclinical evidence that OBP-301 is synergistic with anti-PD-I therapy (**Figure 2**), providing the rationale for this proposal.

Specifically, in a murine model of pancreas and colon cancer, the combination of PD-I inhibition with the murine equivalent of OBP-301 (OBP-502), the combination therapy was associated with immunogenic cell death<sup>48</sup>. OBP-502 induced a significant accumulation of tumor infiltrating lymphocytes within the tumors compared with control. The combination of OBP-502 and PD-I Ab significantly suppressed CT26 colon cancer subcutaneous tumors and successfully eradicated 4/12 (33% of mice. When these 4 tumor-free mice were rechallenged by inoculation with CT26 colon cancer cells, 2/4 (50%) remained tumor free, indicating continued immune surveillance<sup>48</sup>. (Figure 4)



Figure 4 Antitumor activity of the combination of OBP-502 in combination with PD-I Ab inhibitor. (A) study schema, CT26 and PAN02 are murine colon and pancreatic tumor models. OBP-and PDIAb were administered 3 times as indicated. (B) Tumor growth curves with control PD-I Ab, OBP-502: or the combination

The optimal treatment for human cancer requires a therapeutic ratio that increases cytopathic efficacy to target tumor cells, rather than surrounding normal cells. Thus, focus on the genetic and epigenetic targets present only in cancer cells is providing an expanding repertoire of clinically applicable targeted therapeutics, including the use of oncolytic viral vectors.

Oncolytic immunotherapy employs viruses that are designed to preferentially replicate in and lyse cancer cells and through this process trigger antitumor immunity. Following the first description of a virus engineered to replicate selectively in cancer cells over 20 years ago, the field of oncolytic immunotherapy has expanded dramatically. Over 10 different viral species have now been assessed or are under assessment in human studies, including the oncolytic virus-based product (Onyx-015 adenovirus), which entered a Phase III clinical trial in the United States (US), and a similar virus, H101, which was approved for use in combination with chemotherapy as a treatment for Head and Neck cancer by the Chinese State Food and Drug Administration in November 2005. More recently, a Phase III pivotal trial of *talimogene laherparepvec* (T-VEC), an oncolytic herpes virus expressing granulocyte-macrophage colony stimulating factor (GM-CSF) in patients with advanced melanoma met its primary endpoint, demonstrating a significant improvement in durable response rate versus GM-CSF alone (16% vs 20%, p<0.0001) 49. Based on these results, in October 2015, IMLYGIC (talimogene laherparepvec) was granted approval as the first oncolytic viral therapy in the US indicated for the Local Treatment of Unresectable Cutaneous, Subcutaneous and Nodal Lesions in Patients With Melanoma Recurrent After Initial Surgery<sup>50</sup>. The European Medicines Agency also recommended authorizing Imlygic for the treatment of adults with unresectable melanoma that is regionally or distantly metastatic (Stage IIIB, IIIC and IVM1a) with no bone, brain, lung or other visceral disease<sup>51</sup>.

Conditionally replicative oncolytic viruses (CRAds) are engineered for selective replication in cancer cells that express certain oncogenic phenotypes<sup>52-53</sup> To this end, multiple viral backbones have been employed, although the most commonly utilized is derived from the adenovirus serotype 5 (Ad5). OBP-301 is a novel, replication-competent Ad5-based adenoviral construct that incorporates a human telomerase reverse transcriptase gene (hTERT) promoter (Figure 5). The hTERT promoter encodes for the catalytic protein subunit of telomerase, a polymerase that acts to stabilize telomere lengths and is highly expressed in tumors but not in normal, differentiated adult cells. The adenoviral reproductive cycle is a highly orchestrated process. At the molecular level, the adenoviral genome contains 8 transcriptional units that are activated at different phases of infection. They are referred to as early (EIA), immediate early (EIB, E2, E3, E4), intermediate (IX and IVa2), and late genes. In the construct of OBP-301, the normal transcriptional regulatory element of the EIA gene is replaced by the hTERT promoter and additional modifications to enhance specificity include the replacement of the normal transcriptional element of viral E1B gene by an internal ribosomal entry site (IRES) sequence to minimize "leakiness". In the resulting replication-selective, tumor specific adenovirus vector OBP-301, the hTERT promoter element drives the expression of E1A and E1B genes linked with an internal ribosome entry site. Furthermore, OBP-301 is the first replication-competent adenovirus that retains a fully functional viral E3 region, which codes for proteins that regulate the immune response to the virally infected cel152.

## OBP-301 (Telomelysin)



AE I = delta El adenovirus vector, E IA, E 1B = transcriptional units, hTERT = human telomerase reverse transcriptase, RES = internal ribosomal entry Site, ITR = inverted terminal repeat

## Figure 5 The construct of OBP-301

OBP-301 construct is taken by the cells expressing the Coxackie Adenovirus Receptor (CAR). It has been shown by Oncolys researchers that radiotherapy upregulates the expression of this receptor on the surface of tumor cells. Once the virus reaches the nucleosome it remains episomal

because there is no homology between the virus genome and the host genome. Important note: After entering the nucleus, the DNA of the virus does not integrate in the host DNA: it always remains episomal. This is a safety feature of Adenoviruses as a class that makes them attractive therapeutic constructs <sup>20, 66</sup>. Specificity to cancer is derived by exploiting differential (normal versus tumor) cell surface or intracellular aberrations in gene expression that arise in malignancies. Telomerase activation is considered to be a critical step in carcinogenesis, and its activity is closely correlated with hTERT expression. Thus, expression of hTERT is generally low in differentiated adult cells, and active in cells with proliferative capacity such as tumors, gastrointestinal endothelium, or stem cells <sup>24, 53</sup> with the majority of malignant tumors shown to demonstrate high telomerase activity. Previous studies have demonstrated control over the expression of exogenous genes to telomerase-positive cancer cells by the hTERT promoter <sup>54</sup> and the hTERT promoter is an excellent candidate for generating cancer-specific oncolytic adenovirus.

There are several mechanisms by which adenoviruses in general, and OBP-301 in particular, can destroy tumor cells *in vivo*. Direct cell lysis occurs following viral replication and data from animal models have shown that non-replicating adenovirus in rodent tissue will induce both an acute (2-4 days) and chronic (14 days) inflammatory infiltration. During the acute phase, tumor necrosis factor (TNF-a) and interleukin (IL)-1 and IL-6 are produced in high concentrations locally within the tissue. These cytokines have both direct cytopathic effects and indirect effects through immune effector cell recruitment into the local tissue. Finally, adenovirus infection of a tumor cell may augment tumor antigen presentation and enhance tumor antigenicity, leading in turn to improved recognition and destruction of tumors by cytotoxic T cells.

*In vitro* studies have validated the selective infectivity and direct cytolysis of OBP-301 in cancer cells and *in vivo*, intratumoral injection has demonstrated anti-tumor activity without significant toxicity. Additionally, distant viral uptake was observed following intratumoral injection, evidenced by the presence of adenoviral protein in non-injected tumors following treatment of the contralateral tumor. These encouraging pre-clinical findings of safety and directed antitumor activity were supportive of the continuing clinical development of OBP-301 as an oncolytic therapeutic agent.

### 1.4 Summary of Non-Clinical and Clinical Studies

#### 1.4.1 Non-Clinical Studies

The pre-clinical experience with OBP-301 is described in further detail in the Investigator's Brochure<sup>55</sup>. Non-clinical studies have investigated OBP-301 mechanism of action and clinical proof-of-concept in a) cytotoxicity studies using normal and tumor cells, and b) tumor-bearing xenograft mouse models. The safety of OBP-301 has been characterized in animal models that exhibit tumors (xenograft models) as well as in non-tumor models (normal cotton rats, *Sigmodon hispidus*). The primary safety studies for OBP-301 were conducted in cotton rats, a species selected based on information available in the literature, which suggested that this was a relevant and semi- permissive model for adenoviral safety characterization and reflecting a

pre-investigational new drug application (pre-IND) discussion with the Center for Biologics Evaluation and Research (CBER) at the US Food and Drug Administration (FDA).

Due to issues with the generation of homologous recombinants when using an human embryonic kidney cell (HEK) 293 cell substrate for OBP-301 manufacture, transfer to a HeLa cell-based production system was implemented after pre-clinical studies had been initiated. The HEK293 cell-based material may have contained wild-type Ad5, which may have contributed to the observed oncolytic activity. Comparability studies undertaken m the rodent toxicology species, consisting of extended product characterization and a comparison of the toxicological effect of the HEK293 and HeLa OBP-301 material, have demonstrated equivalence between OBP-301 virus produced through either production system.

## Non-clinical Pharmacology

In vitro studies have demonstrated cytopathic activity of OBP-301 on a variety of human tumor cell lines derived from different organs relevant to the clinical setting, as evaluated by a cell viability assay (XTT assay). OBP-301 oncolytic activity in tumor cells was found to be similar compared to another engineered oncolytic virus, and was similar to or slightly weaker than that of wild-type Ad-5 depending on the target tumor cell type. Cytopathic activity of OBP-301 in human normal cell lines was also evaluated, using a variety of methods (XTT assay, plaque assay, Coomassie Blue staining), including assays for E1A mRNA and protein expression, which served as surrogates for viral replication. A correlation between the expression of E1A, hTERT activity and viral replication at the early stage of infection appeared to be present. In normal cells, OBP-301 is less cytotoxic than wild-type Ad5, while in tumor cell lines, OBP-301 showed cytopathic effects equivalent to wild-type Ad5. This is indicative of selective replication in the tumor cells.

In mechanism-of-action studies, there appeared to be a correlation between E1A expression (assessed by immunoblot) and hTERT mRNA expression levels in tumor cells at the early stage of infection. In addition, a correlation between Coxsackie adenovirus receptor (CAR) expression and cytopathic effect of OBP-301 was noted for tumor cells. *In vivo*, the human tumor-bearing xenograft mouse model was utilized in order to define a potentially efficacious dose and regimen. In the first study, multiple intratumoral injections of OBP-301 E3 (-) and E3 (+) both resulted in equivalent inhibition of tumor growth. A second study demonstrated OBP-301 replication in non-injected distant tumors, as evaluated by RT-PCR for E1A mRNA and immunohistochemistry using an anti-E1A antibody, indicating the potential for OBP-301 to reach and then replicate in distally located tumors. The dose of  $3.6 \times 10^9$  viral particles (VP)/animal intratumoral injection in the xenograft model achieved the anticipated anti-tumor effect, and no drug-related death has been observed.

#### Toxicology

In total, 4 single dosing toxicological studies with OBP-301, including 2 single non-Good Laboratory Practice (GLP) study and 2 GLP studies, have been undertaken. Most of the data gathered from non-GLP and GLP studies assessed the route in animals most similar to human intratumoral dosing, being the intramuscular (IM) route. Toxicity evaluation following IM

injection of OBP-301 in rats did not show a formal no effect level (NOEL). However, the low dose group,  $10^9$  VP/animal (approximately  $10^{10}$  VP/kg) showed only sporadic, minimal-to-mild, transient microscopic changes in the liver on Day 28, and these changes were no longer apparent by day 85 after treatment. Therefore, this dose was designated to be the No Adverse Effect Level (NOAEL). A higher IM dose,  $10^{11}$  VP/kg (dose group 3 in FXT00014) as well as the highest dose, showed minimal-to-mild sporadic hepatocellular damage on histopathological evaluation. No animals experienced morbid changes, weight loss, or deaths when  $10^{11}$  VP/animal (approximately  $10^{12}$  VP/kg) was administered via either the intravenous (IV) or IM route.

In the pilot repeated dose study, rats (15 males and 15 females) were assigned into 3 groups, Group 1: Control group, Group 2: 7 days repeated dosing and Group 3: 14 days repeated dosing. Both groups 2 and 3 had a 7-day Follow-Up Period following the dosing phase. The results of this study demonstrated that repeat dosing of IM administered OBP-301 to cotton rats at  $1 \times 10^{11}$  VP/animal for 7 or 14 day was well tolerated. No significant differences were observed in animals dosed for either 7 or 14 days.

In the single dose toxicity study of intra-hepatic injection, histopathologic findings were observed including adhesion, fibrinous inflammation, granulomatous inflammation, and necrosis in the liver on Day 5 and adhesion and fibrosis in the liver on Day 14 in both genders at  $1 \times 10^{11}$  VP/kg. However, no mortality, or observations of clinical signs, body weight and food consumption changes were reported. Systemic distribution of virus away from the injection site was noted in these studies with quantitative PCR (qPCR) data at 10<sup>11</sup> VP/animal indicating the presence of viral DNA in the liver (and to a lesser extent in the lung) out to and including Day 85. These data showed continued presence of viral DNA in normal liver, which may signify that the toxicity on histopathologic evaluation in the liver was test article related (highest dose only, other dose groups were not evaluated for persistence). However, the continued presence of viral DNA in the highest dose group did not result in accrual of toxicity with lesions identified on Day 85, particularly the liver lesions noted above, no more severe than those observed at earlier time points. In addition, the pattern of persistence was consistent with results from other replication-competent oncolvtic adenoviruses (see December 2005 RAC Meeting Documents Tab 2397, Protocol Number 0510-732: A Phase I/II Dose Escalation Trial of Intratumoral Injection with Oncolytic Adenoviral Vector INGN 007 (VRX-007) in Patients with Advanced Solid Tumors). IM compared to IV administration was shown to limit toxicity, and all toxicities were reflected in the biomarker surrogates of clinical pathology.

Dosing in human patients will utilize a conservative dose extrapolation paradigm and offers an adequate safety margin for systemic toxicity. The human equivalent dose (HED) is calculated on a body weight-adjusted basis (to  $10^{10}$  VP/kg × 70 kg, or  $7 \times 10^{11}$  VP; the HED). The highest proposed clinical dose of  $1 \times 10^{12}$  VP (equivalent to ~1.4 ×  $10^{10}$  VP/kg) is equivalent to the NOAEL dose in the animal studies.

#### 1.4.2 Clinical Studies

Clinical trials of OBP-301 administered by intratumoral injection have been conducted in patients with advanced cancer under the following protocols:

## Completed studies

OBP-301-001: an open-label, Phase I, dose-escalation study. The first human study evaluating sequential doses of a single  $(1 \times 10^{10} \text{ to } 1 \times 10^{12} \text{ VP/tumor})$  and repeated  $(1 \times 10^{12} \text{ VP/tumor})$  intratumoral injection of OBP-301 in patients with advanced solid carcinoma. The first patient was enrolled on 30 October 2006 and the last patient completed follow-up on 24 October 2011. Twenty-two patients (n = 13 female, n = 9male) were treated and analysed. Patients with the following tumor types participated in the Phase 1 trial: 5 patients with melanoma, 4 with squamous cell carcinoma of the head and neck, 3 with breast cancer, 2 with soft-tissue sarcoma, and 1 each with squamous cell carcinoma primary unknown, carcinoma of the salivary gland, non-small cell lung cancer, neuroendocrine tumor, basal cell carcinoma, carcinoma of the gall bladder, pancreatic carcinoma, and cancer of the vulva. Of these, 3 patients (1 patient with carcinoma of the breast and the 2 patients with carcinoma of the gall bladder and pancreatic carcinoma, respectively) had visceral administration of OBP-301, all into the liver. The study was conducted under the current IND for OBP-301. OBP-301 was found to be well tolerated in this Phase I study. No dose-limiting toxicities (DLTs) were experienced by any of the 22 patients treated with OBP-301 in this study; therefore, the maximum tolerated dose (MTD) could not be determined. Analysis of all safety data from this study demonstrated an acceptable safety profile with intratumoral injection of OBP-301 with types of events reported that were similar to those reported in patients receiving other adenovirus vectors. Signals of efficacy were seen even in patients treated with a single intratumoral injection. Most patients had stable disease after treatment (15/17); 2 patients reported progressive disease on Day 28. One additional patient who had stable disease on Day 28 reported progressive disease on Day 56. In patients followed for up to 5 years after study participation, there was no signal of a safety concern related to OBP-301 treatment.

#### Retrospective analyses:

**A.**Biopsy samples were obtained from Case C-S, a 60-year-old black male patient enrolled in the Phase I study, who had a diagnosis of squamous cell carcinoma in mouth (Stage IVa). OBP-301 was injected in the tumor in submandibular area. Tumor shrinkage was observed within 7 weeks after injection. Biopsy samples were obtained from the injected site on Day 28 after injection and evaluated retrospectively for histopathological and immunological responses. Results demonstrated tumor cell degradation accompanied by increased numbers of antigen presenting cells (APC), CD8+ T cells, and a decreased regulatory T cell (T<sub>reg</sub>) population, suggesting treatment-induced oncolysis and immunological activation. In this patient, the anti-tumor effect of OBP-301 appeared to be mediated by direct cytopathic activity following immunological activation.

**B.**Five patients with melanoma were extracted from the total population of patients enrolled in the Phase I study for a retrospective analysis. Changes in tumor size in OBP-301 injected and non-injected lesions, and survival duration were calculated. As for the main study, the effect of treatment on tumor reduction was observed in distant non-injected lesions as well as injected lesions in patients with advanced melanoma.

Furthermore, the median survival time was 31.3 months in 5 patients with melanoma<sup>56</sup>. In other reports, the median overall survival of patients diagnosed with unresectable melanoma in Stage IV M1a, M1b, and M1c, are 22.3 months, 11.2 months and 5.1 months, respectively<sup>57</sup>. Survival in patients with other types of tumor who had been treated in the Phase I study was 8.0 months. The results of this retrospective analysis in a subpopulation of patients were suggestive of a positive anti-tumor effect and extended survival in patients with melanoma treated with OBP-301 compared to other types of tumor and other therapies<sup>56</sup>.

#### Other studies:

A.OBP-301-003-C-V (NCT0321305): a Phase I/II dose-escalation study to determine the safety and efficacy of OBP-301 at doses of  $1 \times 10^{10}$  VP/tumor,  $1 \times 10^{10}$  VP/tumor and  $1 \times 10^{12}$  VP/tumor in patients with head and neck or/and thoracic malignant cancers with radiation therapy is being conducted in Japan under Ministry of Health, Labour and Welfare (MHLW) approval (granted on 13 July 2012). The study was initiated on 29 November 2013 and aims to recruit a maximum of 24 patients from Okayama University Hospital in Japan. The primary objectives are assess the clinical safety of OBP-301 in combination with radiotherapy in patients with head and neck or/and thoracic malignant cancers; to determine the MTD/maximum feasible dose (MFD) of OBP-301 and to assess the DLT of OBP-301. Secondary objectives for this study include determination of the tumor response rate of OBP-301 and the duration of response and overall survival. Thirteen patients with esophageal cancer were enrolled in this study, 12 subjects' histological type were squamous carcinoma and one was adenocarcinoma. The safety was monitored when OBP-301 were administered in the dosing levels of; 1 mL of 1x10<sup>10</sup> VP/mL(Level 1), I mL of 1x10<sup>11</sup> VP/mL(Level 2), and 1mL of 1x10<sup>12</sup> VP/mL (Level 3), 3 times of the administration, with the dose escalation study design. Multiple doses of OBP-301 were well tolerated (1 x10<sup>10</sup>  $\sim$ 1 x10<sup>12</sup> VP/ injection), and no DLT and no any intolerable adverse events was observed. Indication of reduction in area of treated tumor was observed in 11 (8 clinical CR and 3 PR) out of 12 evaluable subjects (objective response rate: 91.7%). Pathological responses were also observed in 8 patients (66.7%).

**B.**TL04001 (NCT03213054): a phase 1 study to evaluate the safety of OBP-301, OBP-301 in combination with radiation therapy in patients with esophageal cancer not applicable for standard therapy. The study aims to recruit a maximum of 12 patients in two sites in Japan. The dose of OBP-301 will be started from 3 x 10<sup>11</sup> VP in Cohort 1, and if no any DLT is observed, dose will be escalated to 3 x 10<sup>12</sup> VP. OBP-301 will be injected to primary tumor by endoscopy at Day 1, Day 18 and Day 32. From Day 4, patients receive 6 weeks radiotherapy (60 Gy total).6 patients were enrolled to the phase I clinical trial, 3 patients were treated with 3 x 10<sup>11</sup> VP and 3 x 10<sup>12</sup> VP of OBP-301 in the Cohort 1 and Cohort 2, respectively. No any DLT was observed in this study, thus MTD of OBP-301 was not determined, and MTD was over 10<sup>12</sup> VP/mL. 4 of 6 patients experienced complete response (CR) in primary tumor and CR rate for primary tumor was 66.7%, and other 2 patients also experienced tumor shrinkage.

C.TL03001: a phase II study to evaluate the efficacy, safety, and immunological response of OBP-301, in patients with unresectable metastatic melanoma. The study aims to recruit a maximum of 50 subjects from 5 clinical sites in the US. The first subject was dosed in July 2017. Four subjects were enrolled into this study and subject enrollment of the study was prematurely discontinued in December 2018 due to poor enrollment. The result of this study is being summarized.

## Ongoing studies

**A.** CT-OT-21 (NCT02293850): a Phase I Study to Evaluate the Safety and Efficacy of OBP-301 at doses of  $1 \times 10^{10}$  VP/subject and  $6 \times 10^{12}$  VP/subject in patients with hepatocellular carcinoma. The study aims to recruit a maximum of 36 patients from 2 clinical trial sites in two countries, Taiwan and Korea. A maximum of 36 patients with hepatocellular carcinoma meeting all inclusion criteria and none of the exclusion criteria will be recruited in the trial. For dosing cohorts of at least 3 patients each are planned to be sequentially accrued until study agent related DLT is met in equal or more than 2 patients at whichever dose level. Recruitment to this study commenced in November 2014. In this study, the safety of more than 2 mL has been investigated. In single dose cohorts, 3mL of  $1 \times 10^{12}$  VP/mL ( $3 \times 10^{12}$  VP) was administered in 3 subjects and no DLT was observed.

- **B**. EPOC1505 (NCT03172819): a phase I study to evaluate the safety and potential efficacy of OBP-301 in combination with pembrolizumab in patients with advanced or metastatic solid tumors. This study aims to recruit a maximum of 28 patients in two sites in Japan. As of November 2019, 19 patients have been enrolled and the study is ongoing.
- C. 1807019403: a phase II study to evaluate the efficacy, safety and immunological response of OBP-301 in combination with Pembrolizumab in patients with advanced or metastatic gastric or gastroesophageal junction adenocarcinoma. This study is an investigator initiated clinical study. This study aims to recruit a maximum of 41 subjects at multiple sites in the US. As of November 2020, 8 patients have been enrolled and the study is ongoing.

#### 3.5 Summary of Potential Risks and Benefits

The side effects listed below are expected based on those seen with the same type of adenovirus-based oncolytic agents in human trials and are anticipated from non-clinical toxicological studies of OBP-301 treatment:

Arthralgia Chills
Dehydration Erythema
Fatigue Headache

Injection Site Reaction (Bruising, Erythema, Pain)

Lymphocyte count decreased

Malaise Musculoskeletal Pain

Myalgia Nausea

Oedema Peripheral Pain in Extremity

Pyrexia Tachycardia Tumor Necrosis Vomiting Skin Inflammation Tumor Haemorrhage Tumor Related Complication

In the Phase I study conducted in patients with advanced cancers (OBP-301-001), intratumoral injection with OBP-301 at dose of  $1 \times 10^{10}$  VP/tumor and  $1 \times 10^{12}$  VP/tumor was well tolerated with no DLTs reported<sup>24</sup>. Five patients reported 9 serious adverse events (SAEs) of dysphagia and difficulty breathing, syncope, intractable pain, ECG T-wave abnormality, abdominal pain, ascites, hypotension, chills and pyrexia. Although only patients in the 2 highest dose cohorts reported SAEs, none of the events occurred in more than one patient. SAEs of chills and pyrexia were considered related to drug treatment whereas the causality of all other SAEs was assigned to tumor progression, prior medical conditions, and/or dehydration. Decreases in lymphocytes were noted at the time of treatment, but these changes were transient and returned to baseline levels by no later than Day 7. The changes were not considered to reflect drug toxicity. No consistent changes were observed in the hematological or biochemical laboratory parameters and there was no indication of hepatic, renal or bone marrow toxicity. In summary, analysis of available safety data from this Phase I study demonstrated an acceptable safety profile for intratumoral injection of OBP-301, which exhibited similar events to those reported in patients receiving comparable adenovirus vectors.

There are no known direct benefits to the participants in this study.

## 3.6 Dosage and Treatment Periods

The OBP-301 NOAEL in a GLP rodent species toxicology study was  $10^9$  VP/animal (approximately  $10^{10}$  VP/kg). Higher doses (> $10^{11}$  VP/kg), administered IM, showed minimal-to-mild sporadic hepatocellular damage on histopathological evaluation but no animals experienced morbid changes, weight loss, or deaths when  $10^{11}$  VP/animal (approximately  $10^{12}$ VP/kg) was administered either via the intravenous (IV) or IM route. Furthermore, administration of  $3.6 \times 10^9$  VP via intratumoral injection in a pre-clinical xenograft model achieved demonstrated oncolytic activity. The HED is calculated on a body weight-adjusted basis (to  $10^{10}$  VP/kg × 70 kg, or  $7 \times 10^{11}$  VP; the HED) with the highest proposed clinical dose in this study,  $1 \times 10^{12}$  VP (equivalent to  $\sim 1.4 \times 10^{10}$  VP/kg), equivalent to the NOAEL dose in the animal studies. In the Phase I study in patients with advanced solid carcinoma, the starting dose was a single intratumoral injection of  $1 \times 10^{10}$  VP ( $1.4 \times 10^8$  VP/kg) per tumor. This was administered to an initial 3 cohorts (n = 3 each) and escalated to a maximum of  $5 \times 10^{12}$  VP/tumor. As DLT was not observed with single injections of the highest dose, a repeat dose ( $5 \times 1 \times 10^{12}$  VP), was administered. No DLTs were reported in this patient population with the dosing regimen described.

#### 3.7 Patient Population

Patients with locally advanced head and neck cancer that are not eligible for salvage surgery will be included. Subjects must have already received chemoradiation in combination using a platinum-based chemotherapy and are immunotherapy naïve.
#### 4 OBJECTIVES

# **Primary Objective:**

- To examine the ORR of OBP-301 in combination with pembrolizumab and SBRT in advanced head and neck squamous cell cancer as assessed by the RECIST 1.1 response rate.
- To evaluate the safety of the combination of multiple intratumoral injections of OBP-301 with SBRT and pembrolizumab.

# **Secondary Objectives:**

To evaluate:

- Overall survival (OS) at 1 year.
- Progression free survival (PFS).
- Disease control rate at 6 months.
- Immune related Response Rate (irRR).
- Time to response in non-target lesions.

# **Exploratory Objectives (optional):**

- To determine viral related biomarkers in the tumor: i.e. proof of the presence of the replicating virus (i.e- Adenovirus Hexon Protein) in the tumoral tissue or/and presence of the receptor for Coxsackie Adenovirus Receptor (CAR).
- To examine the tumor-immune microenvironment prior to and following OBP-301, SBRT and pembrolizumab therapy.
- To examine treatment response to OBP-301 + SBRT + pembrolizumab by monitoring changes in plasma and tumor-tissue exosomes and circulating tumoral DNA.
- To examine and characterize the intra-tumoral and systemic immune responses by multi-parameter flow cytometry.
- To determine changes in circulating tumor cells as quantified by the TelomeScan, a liquid Biopsy diagnostic tool. The blood of 10 patients at a maximum of 4 time points will be analyzed.

#### 5 STUDY DESIGN

# 5.1 Study Overview

This is a phase II study of OBP-301 with pembrolizumab and SBRT in recurrent inoperable head and neck cancer that has progressed after initial surgery and/or chemoradiation for advanced disease. The efficacy of pembrolizumab monotherapy is modest in second or third line of treatment of advanced head and neck cancer (~response rate 22%). SBRT reirradiation in patients that received prior surgery and chemoradiation for advanced disease is associated with a response rate

of approximately 60% and with approximately 30-50% 1-year survival. This study will examine the addition of OBP-301 with pembrolizumab and SBRT in patients with recurrent inoperable head and neck cancer that has progressed after initial surgery and/or chemoradiation for advanced disease.

The study schema is provided in Fig 6.



Figure 6 Study Schema

A total of up to 36 patients will be enrolled in a two stage parallel cohort design.

Enrollment will proceed in two stages in each cohort:

• In the first stage, 12 patients will enter the study, if 8 or more patients respond, enrollment will be extended to 36 patients.

The plan is to inject the tumor(s) with OBP-301, if tolerated and no progression, up to twelve injections in each patient.

- All patients will receive OBP-301 at a concentration of  $1 \times 10^{12}$  VP/mL.
- Patients will be able to receive up to a total of  $4 \times 10^{12}$  VP depending on the size of the target tumors (see dosing section 5.2.2 below).
- If the targeted injected lesion disappears, another lesion can be selected for injection.

Study treatment schedule will consist of the following [refer to Figure 6]:

The tumor will be injected with OBP-301 alone at D1. At D8 patients will received intratumoral OBP-301 and systemic pembrolizumab. Radiotherapy with SBRT and OBP-301 injections will start at D15. Intratumoral OBP-301 and systemic pembrolizumab will be started again one week after the 5<sup>th</sup> dose of SBRT at D36 initially for additional 9 doses of the combination OBP-301-pembrolizumab (up to 12 doses of OBP-301 administered) then pembrolizumab alone will be administered systemically for up to 1 year.

#### Of note:

- 1. All the lesions will be irradiated.
- 2. In order to observe a potential response in the non-injected lesions, if several tumors are present, biopsies will be taken at baseline (Day 1) and on Day 18 both from an injected tumor and a non-injected tumor and a comparison will be done between them.
- 3. Standard fine needle biopsies will be taken on the following days:
  - 1) Day 1, prior to therapy.
  - 2) Day 8, prior to therapy (to see the effect of OBP-301 alone),
  - 3) Day 18, prior to therapy (to see the effect of OBP-301 together with pembrolizumab) Given the fact that three biopsies will be done within approximately 3 weeks and special attention will be given to potential side effects (i.e. bleeding, etc.) that can be associated with the biopsy procedures.
  - 4) Optional on Day 94 +/- 5 days (to see the effect of OBP-301 + pembrolizumab + SBRT).

# **6 STUDY POPULATION**

#### **6.1** Selection of Study Population

Only those patients will be included in the study that meet inclusion and exclusion criteria as outlined below.

#### 6.2 Inclusion Criteria

Patients who meet all of the following criteria will be considered for inclusion in the study:

# **Inclusion Criteria:**

Patients who meet all of the following criteria will be considered for inclusion in the study:

- 1. Be willing and able to provide written informed consent/assent for the trial.
- 2. Be  $\geq$ 18 years of age on the day of signing the informed consent.
- 3. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

- 4. Have histologically or cytologically confirmed advanced head and neck squamous cell cancer with cutaneous, subcutaneous or nodal tumors deemed as injectable lesions [see definition below] and have measurable disease for the primary study endpoint of overall response rate by RECIST 1.1 and iRECIST. In addition they must have:
  - 4.1. A single measurable tumor at least 1 cm in size and amenable to intratumoral injection or
  - 4.2. Multiple measurable tumors that in aggregate have a longest diameter of  $\geq 10$  mm

# Note: Injectable lesion definitions: lesions amenable to percutaneous approach, if technically feasible

- 5. Recurrent and inoperable tumor, progressing after prior radiation with curative-intent for advanced disease (adjuvant or definitive with or without chemotherapy or cetuximab). No prior treatment for local regional recurrence (LRR).
- 6. Tumor may be either HPV+ or HPV-.
- 7. Tumor must be PD-L1 positive, defined as CPS  $\geq 1$ .
- 8. Be willing to provide tissue; newly obtained biopsy specimens or formalin-fixed, paraffin-embedded (FFPE) block specimens.
- 9. Female subjects of childbearing potential have a negative urine or serum pregnancy test within 14 days prior to enrollment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. It is permissable that this serum test be performed on the same day as the urine pregnancy test; no more than 14 days prior to enrollment. And male / female subjects of childbearing potential must agree to use an adequate method of contraception starting with signing the informed consent through 120 days after the last dose of study medication.
- 10. Demonstrated adequate organ function as defined in following criteria. All screening labs should be performed within 14 days of enrollment. Note: Subject must not have taken transfusion, hematopoietic agent; granulocyte-colony stimulating factor (G-CSF) etc., and/or oxygen supplementation within 7 days before the screening labs.
  - A) Absolute neutrophil count (ANC)  $\geq 1,000 \text{ /mm}$ 3
  - B) Platelets  $\geq 100,000 \text{ /mm}$ 3
  - C) Hemoglobin  $\geq 9.0 \text{ g/dL}$
  - D) Serum total bilirubin  $\leq 2.0 \text{ mg/dL}$
  - E) Aspartate aminotransferase (AST) (SGOT) and alanine aminotransferase (ALT)  $(SGPT) \le 2.5x$  Upper limit of normal (ULN). For subjects with liver metastases  $\le 5x$  ULN.
  - F) Serum creatinine ≤ 1.5 mg/dL; or if serum creatinine >1.5 mg/dL, measured or calculated creatinine/clearance ≥ 60 mL/min (Cockcroft-Gault formula).
- 11. Life expectancy of  $\geq 6$  months from the first OBP-301 treatment.
- 12. Understand the study requirements and the treatment procedures, and is willing to comply with all specified follow- up evaluations, and provides written informed consent before any study-specific tests or procedures are performed

#### 6.3 Exclusion criteria

The presence of any of the following criteria will exclude the patient from the study:

#### **Exclusion Criteria:**

The presence of any of the following criteria will constitute cause for the exclusion of the participant:

- 1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 2 weeks (chemotherapy, small molecule), or 3 weeks (antibody) of study Day 1.
- 2. Has an active autoimmune disease that has required systemic treatment in past 2 years.
- 3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (greater than the equivalent of prednisone 20 mg/day) or any other form of immunosuppressive therapy within 7 days prior to study Day 1. Daily dose of maintenance prednisone 10mg or equivalent is allowable.
- 4. Has a known additional malignancy that is progressing or requires active treatment, with the exception of stable/low grade tumors that are not expected to influence life-expectancy (e.g. skin SCC, basal cell, differentiated thyroid cancer, prostate cancer on hormonal therapy).
- 5. Has received a live vaccine within 30 days of planned start of study therapy.
- 6. Has a known history of Human Immunodeficiency Virus.
- 7. Has known active Hepatitis B or Hepatitis C.
- 8. Has known history of, or any evidence of active, non-infectious pneumonitis.
- 9. Has an active infection requiring systemic therapy.
- 10. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
- 11. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
- 12. Previous severe hypersensitivity to another monoclonal antibody
- 13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
- 14. Prior intolerance related to severe (≥grade 3) irAE to a prior anti-immune checkpoint inhibitor agent leading to discontinuation of anti-immune checkpoint inhibitor therapy
- 15. Any disorder or condition, or any medication that would put the patient at risk from bleeding after direct tumor injection.
- 16. Not a candidate for SBRT (or equivalent) given for potentially curative intent. All tumors must receive SBRT (or equivalent). For example, patients with locoregional neck recurrence without significant overlap with the previous radiation field, and who do not warrant SBRT for re-irradiation as per the treating radiation oncologist (e.g. out-of-field recurrence), will not be included in the study.
- 17. Received prior immunotherapy with checkpoint inhibitors or other immunotherapy agents.

- 18. Exclude injection of study agent adjacent to great vessels
- 19. Exclude injection into tumor impinging tracheostomy sites
- 20. Exclude subjects with a history of bleeding diathesis
- 21. Exclude patients with abnormal coagulation profile (PT/PTT).
- 22. Exclude subjects that have been treated with two or more courses of radiation therapy to the head and neck, including patients who previously received palliative reirradiation for recurrence.

# **6.3.1 Patient Registration – Part 1 (WCMC Only)**

Patients will be centrally registered with the Office of Billing Compliance. To register a patient, submit the following documents via the JIRA Registration Process:

- Legible copy of the HRBAF
- First and last page of signed informed consent form

Registration must be completed within 24 hours of the signing of informed consent.

# **6.3.2 Patient Registration – Part 2 (All Sites)**

Study participants will be centrally registered Monday through Friday from 9:00am to 4:00pm with the Weill Cornell Medicine Joint Clinical Trials Office (JCTO). To register a new study subject, email the following documents to JCTOIIT@med.cornell.edu:

- Completed WCM subject registration form
- First and last page of the fully executed informed consent form, plus additional pages if checkboxes for correlative studies are required
- Fully executed HIPAA research authorization form
- Eligibility checklist signed and dated by investigator and research nurse
- Documentation of any eligibility waivers granted
- Redacted source documentation to verify eligibility

Note that attachments larger than 4.5 MB are not accepted, so larger attachments should be split into more than one email. Central registration information is reviewed and entered into the REDCap database.

### 6.4 Stopping Criteria

# 6.4.1 Patient Withdrawal Criteria

In accordance with applicable regulations, a participant has the right to withdraw from the study, at any time and for any reason, without prejudice to his future medical care.

Withdrawal from the study and therapeutic measures taken shall be at the discretion of the Investigator. A full explanation for the discontinuation from the study should be made in the participant's medical records and in the eCRF.

Premature discontinuation from active study participation may occur at any time due to any of the following reasons:

- Any situation where, in the opinion of the Investigator or the Medical Monitor, continued participation in the study would not be in the best interest of the patient.
- Positive pregnancy test (see Section for procedures to be followed in case of a pregnancy).
- Patient initiates other anti-cancer therapy. The anti-cancer therapy will be documented in the medical record and eCRF.
- Patient is unable or unwilling to comply with study procedures.
- Patient is lost to follow-up.
- Patient withdraws consent.
- Request by a Health Authority.
- Termination of the study by the study investigator(s).
- Progressive neoplastic disease, unless the Investigator feels this may be pseudoprogression, in which case the patient may remain on study until the next evaluation for extent of disease.

The reason(s) for premature study discontinuation/withdrawal should be reported in the eCRF and within the source documents along with the date of withdrawal. AEs should be documented according to Section 7.0 Adverse Events.

For all patients who discontinue, a Final Visit will be performed within  $28 \pm 5$  days after the last IP administration. If a participant is withdrawn because of an AE, the Investigator must arrange for the participant to have appropriate follow-up care until the AE is resolved or has stabilized. Unresolved AEs will be followed until the last scheduled follow-up visit or until the Investigator determines that further follow-up is no longer indicated. Investigators should attempt to collect the survival information as dictated in section 6.1.3.

Patients who discontinue the active study participation will not be replaced.

Any enrolled patients who are discontinued before study dosing will be documented as screen failures in the eCRF and replaced. No follow-up is required for these patients.

# **6.4.2** Termination or Suspension of the Study

The drug manufacture (Oncolys BioPharma), Investigator and the IEC/IRB reserve the right to terminate or suspend the study at any time for medical, safety, regulatory, administrative, or other reasons consistent with applicable laws, regulations, and Good Clinical Practice (GCP); however, this should be discussed between the relevant parties beforehand and the reason for such decision recorded. Should this occur, all data available will also be recorded in the eCRFs. The Investigator should notify the IEC/IRB in writing of the study's completion or early discontinuation.

We have included adverse events stopping rule (see Section 8.7.9).

In the event that the study is terminated early, the Investigator should make every effort to follow AEs and SAEs for all patients until the end of the defined follow-up period resolution, until the condition stabilizes, until the event is in the opinion of the Investigator stabilized or determined to be chronic, or until the participant dies or is lost to follow-up. SAEs that occur after the Final Visit, that are thought to be related to the administration of OBP-301, should be reported to Oncolys BioPharma Inc. or designee.

#### 7 STUDY TREATMENTS

# 7.1 Investigational Product (IP) Identification

The OBP-301 clinical study material and product is generated according to current Good Manufacturing Practice (cGMP). Table 1 shows an overview of OBP-301. OBP-301 will be provided by Oncolys BioPharma Inc.

**Table 1** Investigational Product Information

| Investigational product code: | OBP-301 |
|---|---|
| Content: | 2 mL/vial (1×10 <sup>12</sup> VP/mL) |
| Dosage form: | Solution; formulated in 20 mM Tris pH 8.0, 25 mM NaCl with 2.5% glycerin, USP by volume, filled in each 5 mL glass vial |
| Storage method for the investigational product: | Store at ≤ -60°C |

#### 7.2 Dosage and Treatment

- 1. OBP-301 1x10<sup>12</sup> to 4 x10<sup>12</sup> viral particles/treatment day/subject injection as outlined below:
  - Up to a total of 12 total tumor injections may be considered in discussion with the PI (Dr. Doru Paul) which may be given in combination with pembrolizumab after completion of SBRT treatment.
  - Primary tumors that are greater than 5 cm may be administered up to  $4 \times 10^{12}$  viral particles/ subject during the same procedure.
  - For smaller tumors (1.0 -2.5cm and 2.5-5.0cm), 1 ml or 2ml OBP-301 will be injected, accordingly based on the safety as determined by the

ENT surgeon. OBP-301 can be administered to more than one lesion simultaneously.

- 2. Pembrolizumab 200 mg intravenous as per study schedule day 8-36 and then every 3 weeks until disease progression as per study schedule.
- 2. Radiation therapy in the form of Stereotactic Body Radiation Therapy [SBRT] will be given for a total of 5 doses over a period of ten days.

# 7.3 Investigational product

# 73.1 Study Supplies OBP-301

Pembrolizumab will be supplied by commercial vendors.

Oncolys BioPharma Inc. will be responsible for the preparation and labelling of the Investigational Product (IP) in accordance with local regulatory requirements. Oncolys BioPharma Inc. will also provide details of batch numbers and all associated safety and stability data.

Oncolys BioPharma Inc. will be responsible for packaging and shipment of the IP to the site(s). Due to product specific requirements, shipments of IP will be made on dry ice using a validated container and temperature monitoring. An official shipping form to be completed by the study Investigator or designee (e.g., pharmacist) will be included in each shipment. Specific ordering information will be provided to each participating site upon study activation.

# 7.3.1.1 Storage Conditions

The study Investigator or designee is responsible for receiving each shipment of IP. Upon receipt of the IPs at the investigational site, the receipt procedures should be completed and IPs stored appropriately  $\leq$  -60°C. A record to account for all dispensing and return of unused IPs will be maintained by the investigational sites. At the end of the study the IPs will be reconciled. The Investigator will be fully responsible for the security, accessibility, and storage of the IPs while they are at the investigational facility.

Vials must be stored in the original vial storage boxes to facilitate supply tracking. It is recommended to leave the vial storage boxes in the original leak-proof bag or in a substitute leak-proof container, particularly if the supplies are not segregated (i.e., in a separate section of the freezer) from other products or biological samples.

The freezer should be in a locked or secured area, with limited access. Additionally, the freezer should have a temperature recorder and an alarm system. The temperature plot should be properly maintained and checked. Documentation for calibration of the freezer at installation and at each maintenance inspection should be available (at least annually or as per manufacturer's recommendations). A biohazard symbol should be affixed to the outside of the storage compartment.

# 7.3.1.2 Accountability and Compliance

The Investigator, pharmacist, or designee may only dispense clinical supplies in accordance with this protocol.

The Investigator, pharmacist, or designee, is responsible for maintaining an accurate and current record of all clinical supplies received from Oncolys BioPharma Inc., dispensed to the Investigator or destroyed. Accountability records must be maintained throughout the course of the study, showing receipt and disposition of the clinical supplies.

At the end of the study, it must be possible to reconcile delivery records with that of used, unused and destroyed clinical supplies.

The Investigator is also responsible for the education of study staff in the correct administration of the IP.

Additional measures to ensure treatment compliance are not required because the IP will be prepared and administered by study personnel (see Section 7.3.1.3).

# 7.3.1.3 Study Material Preparation

OBP-301 should be prepared according to Biosafety Level 2 Guidelines, unless local regulations require a more rigorous containment level. An outline of Biosafety Level 2 precautions is located in the OBP-301 Pharmacy Brochure Appendix V: Handling Guidelines/Universal Precautions for Biosafety Level 2 Agents. Aseptic technique must be followed at all times during the preparation and transport of the IP to the treatment area. A disinfectant that has been qualified as an effective virucide for adenoviruses should be used for any decontamination procedure. The recommended exposure time should be at least 5 to 15 minutes. However, if the handling precautions recommended by the manufacturer differ, the manufacturer's instructions should be followed.

The duration that the IP remains at room temperature should be minimized and it is recommended that OBP-301 be administered as soon as possible (within 4 hours) after reconstitution. Immediately before injection, the IP may be warmed by rolling the syringe between the palms of the hands, which may facilitate comfort of administration to the patient.

The Investigator is responsible for the education of study staff in the correct administration of the IP and a designated staff member experienced in the administration of investigational agents directly into tumor lesions will administer all treatments.

#### 7.3.1.4 Destruction of Used and Unused Investigational Product

Immediately after use, the used vials should be placed in a biohazardous waste container. Empty or partially used vials should be destroyed, by the study pharmacy, in accordance with institutional biosafety policy and procedures for biohazardous waste management. Proper accounting of the vials must be performed immediately using the Drug Accountability Form.

Written authorization must be obtained from Oncolys BioPharma Inc. before any destruction of unused clinical material supplies. This will occur at the completion of the clinical study or when the expiration date has been reached and could not be prolonged by Oncolys BioPharma Inc. based on updated stability information. In addition, destruction of unused supplies may only be performed after product reconciliation by the monitor.

The unused vials must be destroyed by the study pharmacy, in accordance with institutional Biosafety policy and procedures for biohazardous waste management or returned to Oncolys BioPharma Inc.

The Investigator or designee must fill in, sign, and date the appropriate section of Clinical Trial Material Destruction Certificate. Discrepancies in vial accountability must be explained in writing by the Investigator or designee. A copy will be retained for the site study file and the monitor will retrieve the original.

Further information of the storage, preparation, and administration of IP will be provided in the OBP-301 Pharmacy Brochure.

# 7.3.2 Selection and Timing and IT Administration for each Patient

OBP-301 ( $1\times10^{12}$  VP/mL) is administered as intratumoral injection into a head and neck cancer tumor mass that is suitable for injection, eg greater than 1 cm in size and in a location amenable for injection. The largest diameter of the lesion will determine the volume of OBP-301 injected. Lesions 1-2.5 cm will be injected with up to 1 ml ( $1\times10^{12}$  VP), lesions between 2.6 cm to 5.0 cm in size will be injected with up to 2 ml ( $2\times10^{12}$  VP) and lesions >5cm in size will be injected with up to 4ml ( $4\times10^{12}$ VP). The rationale for this is to ensure adequate penetration of the viral particles throughout the tumor.

Pre-injection planning is the key to success; therefore, a sketch of the tumor and the planned injection sites should be made. The sketch will be helpful in determining the total quantity of study drug to inject.

The tumor to be injected should be  $\ge 1$  cm in length and can be mapped into (preferably at least) 12 sections. The dose (volume) delivered to the lesion(s) (if patient has 2 or more lesions several lesions can be injected) should be within the range of 1.0 to 2.0 mL (Table 1).

For example, in a 3 cm tumor, a total volume of 2 ml (i.e.  $(2x10^{12} \text{ VP})$ ) will be injected in the tumor.

**Table 1: IT administration Volume Guidelines** 

| Lesion Size | Injection Volume |
|--------------------|------------------|
| > 5.0 cm | Up to 4 mL |
| > 2.5 cm to 5.0 cm | 2 mL |

| > 1.0 cm to 2.5 cm | 1 mL |
|--------------------|------|

Note: If lesion shrinks, adjust injection volume according to the lesion size in the table above.

If the tumor disappears, and there are other lesion(s) amenable for injections they should be injected.

# Safety Guidelines for Clinical Study Patients and Caregivers

- Avoid direct contact with body fluids of patients who were injected with OBP-301.
- Immunocompromised individuals or pregnant women should not come into direct contact with body fluids of treated patients.

# Safety Guidelines for Healthcare Staff when Handling OBP-301

- Immunocompromised individuals or pregnant women should not prepare or administer OBP-301 and should not come into direct contact with OBP-301 injection sites, dressings, or body fluids of treated patients.
- Staff must follow Biosafety Level 2 guidelines by avoiding accidental exposure to OBP-301 and follow the instructions for preparation, administration, and handling of OBP-301.
- Staff must wear personal protective equipment (protective gown or laboratory coat, safety glasses or face shield, and gloves) while preparing or administering OBP-301.
- Cover any exposed wounds before handling OBP-301.
- In the event of an accidental occupational exposure (e.g., through a splash to the eyes or mucous membranes), flush with clean water for at least 15 minutes.
- In the event of exposure to broken skin or needle stick, clean the affected area thoroughly with soap and water and/or a disinfectant.
- Clean all surfaces that may have come in contact with OBP-301 and treat all spills with a virucidal agent such as 1% sodium hypochlorite or 70% isopropyl alcohol and blot using absorbent materials.
- Dispose of all materials that may have come in contact with OBP-301 (e.g., vial, syringe, needle, cotton gauze, gloves, masks, or dressings) as biohazardous waste.

# 7.3.3 Injection Procedures

**7.3.3.1** The optimum technique for injection of a primary tumor is to inject the viral particles circumferentailly around the lesion in 12 tracks. This will ensure that the viral particles will be

maximally penetrated into the lesion. More detailed administration instructions can be found in the Pharmacy Manual (Section 6.5).

ENT surgeons will be eligible to perform the procedure in a level 2 biohazard room. A training video (prepared by Oncolys Biopharma) is available as well.

Procedure will take place in the ENT or Interventional Radiology procedure rooms. Standard sterilization procedures will be used. A standard laryngoscope and needle will be used for the procedure. Guidelines for each injection procedure are provided below.

#### **Pre-Injection**

- Confirmation of eligiblity
- Review of medications
- Abbreviated physical exam and performance status
- Vital signs

# Post-Injection

- Monitor patient for 60-90 minutes for any symptoms of injection site pain, bleeding, nausea. There should be a minimum of 1 hour between injection and pembro administration.
- Vital signs (except weight)

OBP-301 may be associated with injection site pain if administered to dermal lesions. However, pain has not been observed for intralumenal injections previously.

#### **OBP-301**

OBP-301 injection will be delayed for any ongoing Grade 3 toxicity at the time of the next scheduled injection. Patients who require a delay of OBP-301 injection of > 4 weeks (i.e., approximately 6 weeks from the previous injection) due to lack of resolution to Grade 1 toxicity will be discontinued from the study. In this circumstance, the patient will be evaluable for toxicity, but will be replaced (up to the maximum enrollment) for efficacy assessment.

# 7.3.3.2 Patient selection for injection

In order to receive intratumoral (IT) injections, patients must have relatively good performance status (ECOG 0-1) and disease in a site that is considered to be amenable to local injection. Suitable sites for injection include cutaneous and subcutaneous nodules over the scalp, face, neck and upper chest wall. In addition, cervical nodal masses in levels I-VI are frequently accessible to injection. Direct injection into mucosal lesions affecting the oral cavity (lip, buccal mucosa, oral tongue, floor of mouth, palate) and oropharynx (tonsil, base of tongue) is also relatively straightforward

and feasible in many patients. Injection of primary tumors of the larynx and hypopharynx present specific challenges and these sites will not be injected. Most patients with squamous cell cancers of the head and neck who are considered for studies of IT will have previously received relatively high-dose irradiation (in either the radical or adjuvant settings). Injection into irradiated sites is usually safe and feasible, but there are specific concerns around injection into sites that have been irradiated on more than one occasion (i.e. re-irradiated), especially if they lie in close proximity to major blood vessels in the neck. Certainly, it would appear sensible to advise caution when considering IT in sites adjacent to the great vessels of the neck that have received cumulative radiation doses >100 Gy. Such concerns will be amplified in patients with any prior history of bleeding from their tumor or in patients who are taking anti-platelet or anti-thrombotic medications. If such therapy cannot be discontinued safely, these patients should not be routinely considered for IT therapy. Many patients entering clinical trials of IT will have loco-regionally recurrent disease that is sufficiently advanced to require them to have undergone tracheostomy (permanent or temporary) and/or insertion of feeding (nasogastric or percutaneous gastrostomy/jejunostomy) tubes. Such interventions can be extremely beneficial for the patient and may extend opportunities for trial entry to patients who might otherwise not be considered suitable. In particular, in patients with bulky nodal masses and/or mucosal disease involving the oropharynx and laryngo-hypopharynx, the presence of a tracheostomy and/or a feeding tube can allay concerns that inflammation and swelling associated with IT might cause airway compromise or loss of the ability to take oral fluids/nutrition. Nevertheless, caution is advised in patients with disease at or around tracheostomy sites. Direct injection of IT into such sites can be associated with airway compromise if treatment-related inflammation narrows the aperture of the stoma. In addition, marked treatment response with disappearance of disease at the stoma can cause difficult problems with stoma care and can be associated with exposure of great vessels in the neck (with resulting risks of major hemorrhage) and fistula formation with the pharynx/upper esophagus.

## 7.3.3.3 Technical considerations

Intratumoral injections into head and neck sites can pose a number of technical challenges that must be recognized and addressed. Squamous cell cancers have a marked tendency to ulcerate/fungate onto the skin surface, which can result in leakage of injected material through the skin surface during drug administration. This can, in turn, result in variable and unpredictable dosing of injected lesions and has frequently been used as an exclusion criterion in clinical protocols. For larger lesions, however, it is often possible to direct the injection into deeper parts of the lesion and deliver the injected material sufficiently slowly to avoid leakage through the surface of the lesion. Similar concerns exist for lesions that demonstrate fistulation between mucosal and cutaneous surfaces in the head and neck. Again, if the lesions are sufficiently large, it is often possible successfully to inject the deeper aspects of the lesions away from the fistulous tract and avoid leakage and loss of the therapeutic agent.

Similar considerations apply when treating patients with large neck masses that have a substantial cystic or necrotic component. Clearly, in such cases, there is a risk that the therapeutic agent might be delivered into a fluid-filled space within the tumor mass where it is unlikely to mediate the

desired biological effects. In such cases, it is possible to perform injections directly without image-guidance if a definite solid component of the tumor can be identified clinically. If that is not the case, it is usually advisable to perform the injections under ultrasonic guidance to enable targeting of solid, viable parts of the tumor.

Another feature of recurrent cancer in the head and neck region is its tendency to be associated with dense fibrosis. This is most frequently seen in patients who have undergone previous surgery and/or irradiation. In such cases, the precise boundaries of the disease can be difficult to define, even with imaging investigations, and injections may have to be delivered using considerable force to overcome the high interstitial pressure in the target tissues. This can lead to spread of the injection into adjacent tissues away from the tumor-bearing site. In such circumstances, injection under image-guidance (preferably ultrasound) at a slow rate is advised in order to retain the injected material at the desired site.

The greatest challenge is presented by patients with disease close to or involving the great vessels in the neck. As discussed above, specific concerns should arise when patients have disease that encases the carotid artery or its branches to 50% or more of the circumference of the vessel or shows radiological signs of invasion of the media or intima of the vessels. In addition, patients with disease that bridges a tissue plane connecting a major vessel to the skin or a mucosal surface must be considered high-risk for a major hemorrhagic complication. In such cases, a major response can lead to the formation of a sinus tract or fistula to the vessel and this can be associated with catastrophic bleeding. Additional risk factors for bleeding include prior radiation therapy to cumulative doses >100 Gy (achieved in patients who have received re-irradiation) and the presence of active bacterial infection in the neck.

#### 7.4 Pembrolizumab

Pembrolizumab is given at a flat dose of 200 mg IV according to the study schedule. There are no dose modifications to this treatment other than temporary or permanent discontinuation of therapy as detailed below.

Adverse events (both non-serious and serious) associated with pembrolizumab exposure may represent an immunologic etiology. These adverse events may occur shortly after the first dose or several months after the last dose of treatment. Pembrolizumab must be withheld for drug-related toxicities and severe or life-threatening AEs as per Table 2 below. See Section 5.2.2.6 and Events of Clinical Interest Guidance Document for supportive care guidelines, including use of corticosteroids.

**Table 2**. Dose Modification Guidelines for pembrolizumab -Related Adverse Events (as per package insert).

| Toxicity | Hold<br>Treatment<br>For Grade | Timing for Restarting Treatment | Discontinue Subject from Study Treatment |
|---|---|---|---|
| Diarrhea/<br>Colitis | 2-3 | Toxicity resolves to Grade 0-1. | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 4 | Permanently discontinue | Permanently discontinue |
| AST,<br>ALT, or | 2 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose. |
| Increased<br>Bilirubin | 3-4 | Permanently discontinue (see exception below) <sup>1</sup> | Permanently discontinue |
| Type 1<br>diabetes<br>mellitus<br>(if new<br>onset) or<br>Hypergly<br>cemia | T1DM or 3-4 | Hold pembrolizumab for new onset Type 1 diabetes mellitus or Grade 3- 4 hyperglycemia associated with evidence of beta cell failure. | Resume pembrolizumab when patients are clinically and metabolically stable. |
| Hypophy<br>sitis | 2-3 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 4 | Permanently discontinue | Permanently discontinue |
| Hyperthy roidism | 3 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 4 | Permanently discontinue | Permanently discontinue |
| Hypothyr<br>oidism | 2-4 | Therapy with pembrolizumab can be continued while treatment for the thyroid disorder is instituted | Therapy with pembrolizumab can be continued while treatment for the thyroid disorder is instituted. |
| Infusion<br>Reaction | 3-4 | Permanently discontinue | Permanently discontinue |
| Pneumon itis | 2 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 3-4 | Permanently discontinue | Permanently discontinue |

| Toxicity | Hold<br>Treatment<br>For Grade | Timing for Restarting Treatment | Discontinue Subject from Study Treatment |
|---|---|---|---|
| Renal<br>Failure<br>or<br>Nephritis | 2 | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| T ( pinitis | 3-4 | Permanently discontinue | Permanently discontinue |
| All Other Drug- Related Toxicity <sup>2</sup> | 3 or Severe | Toxicity resolves to Grade 0-1 | Toxicity does not resolve within 12 weeks of last dose or inability to reduce corticosteroid to 10 mg or less of prednisone or equivalent per day within 12 weeks. |
| | 4 | Permanently discontinue | Permanently discontinue |

Note: Permanently discontinue for any severe or Grade 3 drug-related AE that recurs or any life-threatening event.

# 7.4.1 General Concomitant Medication and Supportive Care Guidelines

Medications or vaccinations specifically prohibited in the exclusion criteria are not allowed during the ongoing trial. If there is a clinical indication for one of these or other medications or vaccinations specifically prohibited during the trial, discontinuation from trial therapy or vaccination may be required. The investigator should discuss any questions regarding this with the Principal Investigator. The final decision on any supportive therapy or vaccination rests with the investigator and/or the subject's primary physician.

#### **Acceptable Concomitant Medications**

All treatments that the investigator considers necessary for a subject's welfare may be administered at the discretion of the investigator in keeping with the community standards of medical care. All concomitant medication will be recorded on the case report form (CRF) including all prescription, over-the-counter (OTC), herbal supplements, and IV medications and fluids. If changes occur during the trial period, documentation of drug dosage, frequency, route, and date may also be included on the CRF.

All concomitant medications received within 28 days before the first dose of trial treatment and 30 days after the last dose of trial treatment should be recorded.

<sup>&</sup>lt;sup>1</sup> For patients with liver metastasis who begin treatment with Grade 2 AST or ALT, if AST or ALT increases by greater than or equal to 50% relative to baseline and lasts for at least 1 week then patients should be discontinued.

<sup>&</sup>lt;sup>2</sup> Patients with intolerable or persistent Grade 2 drug-related AE may hold study medication at physician discretion. Permanently discontinue study drug for persistent Grade 2 adverse reactions for which treatment with study drug has been held, that do not recover to Grade 0-1 within 12 weeks of the last dose.

**Prohibited Concomitant Medications** 

Subjects are prohibited from receiving the following therapies during the Screening and Treatment Phase (including retreatment for post-complete response relapse) of this trial:

- Antineoplastic systemic chemotherapy or biological therapy
- Immunotherapy not specified in this protocol
- Investigational agents other than OBP-301
- Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, BCG, and typhoid vaccine.
- Systemic glucocorticoids for any purpose other than to modulate symptoms from an event of clinical interest of suspected immunologic etiology. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.

Subjects who, in the assessment by the investigator, require the use of any of the aforementioned treatments for clinical management should be removed from the trial. Subjects may receive other medications that the investigator deems to be medically necessary.

The Exclusion Criteria describe other medications which are prohibited in this trial.

There are no prohibited therapies during the Post-Treatment Follow-up Phase.

#### 7.4.2 Rescue Medications & Supportive Care

Subjects should receive appropriate supportive care measures as deemed necessary by the treating investigator. Suggested supportive care measures for the management of adverse events with potential immunologic etiology are outlined below and in greater detail in the ECI guidance document. Where appropriate, these guidelines include the use of oral or intravenous treatment with corticosteroids as well as additional anti-inflammatory agents if symptoms do not improve with administration of corticosteroids. Note that several courses of steroid tapering may be necessary as symptoms may worsen when the steroid dose is decreased. For each disorder, attempts should be made to rule out other causes such as metastatic disease or bacterial or viral infection, which might require additional supportive care. The treatment guidelines are intended to be applied when the investigator determines the events to be related to pembrolizumab.

Note: if after the evaluation, the event is determined not to be related, the investigator is instructed to follow the ECI reporting guidance but does not need to follow the treatment guidance (as outlined in the ECI guidance document). Refer to Section 5.2.1 for dose modification

It may be necessary to perform conditional procedures such as bronchoscopy, endoscopy, or skin photography as part of evaluation of the event. Suggested conditional procedures, as appropriate, can be found in the ECI guidance document.

#### • Pneumonitis:

- o For **Grade 2 events**, treat with systemic corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- o For **Grade 3-4 events**, immediately treat with intravenous steroids. Administer additional anti-inflammatory measures, as needed.
- Add prophylactic antibiotics for opportunistic infections in the case of prolonged steroid administration.

### • Diarrhea/Colitis:

Subjects should be carefully monitored for signs and symptoms of enterocolitis (such as diarrhea, abdominal pain, blood or mucus in stool, with or without fever) and of bowel perforation (such as peritoneal signs and ileus).

- o All subjects who experience diarrhea/colitis should be advised to drink liberal quantities of clear fluids. If sufficient oral fluid intake is not feasible, fluid and electrolytes should be substituted via IV infusion. For Grade 2 or higher diarrhea, consider GI consultation and endoscopy to confirm or rule out colitis.
- o For **Grade 2 diarrhea/colitis** that persists greater than 3 days, administer oral corticosteroids.
- For **Grade 3 or 4 diarrhea/colitis** that persists > 1 week, treat with intravenous steroids followed by high dose oral steroids.
- When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- Type 1 diabetes mellitus (if new onset, including diabetic ketoacidosis [DKA]) or ≥ Grade 3 Hyperglycemia, if associated with ketosis (ketonuria) or metabolic acidosis (DKA)

# o For **T1DM** or **Grade 3-4** Hyperglycemia

- Insulin replacement therapy is recommended for Type I diabetes mellitus and for Grade 3-4 hyperglycemia associated with metabolic acidosis or ketonuria.
- Evaluate patients with serum glucose and a metabolic panel, urine ketones, glycosylated hemoglobin, and C-peptide.

# • Hypophysitis:

For Grade 2 events, treat with corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
 Replacement of appropriate hormones may be required as the steroid dose is tapered.

o For **Grade 3-4** events, treat with an initial dose of IV corticosteroids followed by oral corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.

0

# Hyperthyroidism or Hypothyroidism:

Thyroid disorders can occur at any time during treatment. Monitor patients for changes in thyroid function (at the start of treatment, periodically during treatment, and as indicated based on clinical evaluation) and for clinical signs and symptoms of thyroid disorders.

- o **Grade 2** hyperthyroidism events (and **Grade 2-4** hypothyroidism):
  - In hyperthyroidism, non-selective beta-blockers (e.g. propranolol) are suggested as initial therapy.
  - In hypothyroidism, thyroid hormone replacement therapy, with levothyroxine or liothyroinine, is indicated per standard of care.
- o **Grade 3-4** hyperthyroidism
  - Treat with an initial dose of IV corticosteroid followed by oral corticosteroids. When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks. Replacement of appropriate hormones may be required as the steroid dose is tapered.

#### • Hepatic:

- o For **Grade 2** events, monitor liver function tests more frequently until returned to baseline values (consider weekly).
  - Treat with IV or oral corticosteroids
- o For **Grade 3-4** events, treat with intravenous corticosteroids for 24 to 48 hours.
- When symptoms improve to Grade 1 or less, a steroid taper should be started and continued over no less than 4 weeks.

# • Renal Failure or Nephritis:

- o For **Grade 2** events, treat with corticosteroids.
- o For **Grade 3-4** events, treat with systemic corticosteroids.
- o When symptoms improve to Grade 1 or less, steroid taper should be started and continued over no less than 4 weeks.
- **Management of Infusion Reactions**: Signs and symptoms usually develop during or shortly after drug infusion and generally resolve completely within 24 hours of completion of infusion.

Table 3 below shows treatment guidelines for subjects who experience an infusion reaction associated with administration of pembrolizumab.

#### **Table 3 Infusion Reaction Treatment Guidelines**

| NCI CTCAE Grade | Treatment | Premedication at subsequent dosing |
|---|---|---|
| Grade 1 Mild reaction; infusion interruption not indicated; intervention not indicated | Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. | None |
| Grade 2 Requires infusion interruption but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics, IV fluids); prophylactic medications indicated for < =24 hrs | Stop Infusion and monitor symptoms. Additional appropriate medical therapy may include but is not limited to: IV fluids Antihistamines NSAIDS Acetaminophen Narcotics Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. If symptoms resolve within one hour of stopping drug infusion, the infusion may be restarted at 50% of the original infusion rate (e.g., from 100 mL/hr to 50 mL/hr). Otherwise dosing will be held until symptoms resolve and the subject should be premedicated for the next scheduled dose. Subjects who develop Grade 2 toxicity despite adequate premedication should be permanently discontinued from further trial treatment administration. | Subject may be premedicated 1.5h (± 30 minutes) prior to infusion of pembrolizumab (MK-3475) with: Diphenhydramine 50 mg po (or equivalent dose of antihistamine). Acetaminophen 500-1000 mg po (or equivalent dose of antipyretic). |
| Grades 3 or 4 | Stop Infusion. | No subsequent dosing |
| Grade 3: Prolonged (i.e., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms | Additional appropriate medical therapy may include but is not limited to: IV fluids Antihistamines | |

| NCI CTCAE Grade | Treatment | Premedication at subsequent dosing |
|---|---|---|
| following initial improvement; hospitalization indicated for other clinical sequelae (e.g., renal impairment, pulmonary infiltrates) Grade 4: Life-threatening; pressor or ventilatory support indicated | NSAIDS Acetaminophen Narcotics Oxygen Pressors Corticosteroids Epinephrine Increase monitoring of vital signs as medically indicated until the subject is deemed medically stable in the opinion of the investigator. Hospitalization may be indicated. Subject is permanently discontinued from further trial treatment | |
| | administration. | |

Appropriate resuscitation equipment should be available in the room and a physician readily available during the period of drug administration.

# 7.5 Radiation therapy

Radiation (SBRT) will begin on Day 8

# **Radiation Therapy Guidelines**

- 1. Treatment approaches will use SBRT (or equivalent).
- 2. Localization requirements: All patients will be immobilized and simulated in the treatment position prior to the start of OBP-301. Immobilization devices using an aquaplast mask is recommended. A contrast enhanced CT with immobilization is recommended for planning. Additional diagnostic imaging may be fused to the contrast enhanced CT simulation at the discretion of the treating physician. For patients who cannot receive a contrast enhanced CT simulation, non-contrast CT simulation images should be fused to diagnostic contrast CT, MRI or PET-CT imaging performed within 30 days of the CT simulation. Slice thickness should be optimally 1-3 mm for SBRT.

Patients must be reproducibly immobilized. Radio-opaque markers may be used whenever possible to delineate the surgical scars, extent of nodal disease, skin involvement, and any gross disease. For SBRT, prior to each treatment, socenter or reference point localization images (anterior/posterior and lateral) should be obtained using a cone beam CT or verification imaging.

- 3. **Target volumes:** Appropriate target volumes will be determined at the time of simulation to treat gross disease and areas of potential microscopic disease as determined by the treating physician. All gross disease above the clavicles should be targeted for SBRT in. Two target volumes will be defined on each CT slice: GTV and PTV. In cases of multiple tumor sites, the treating physician may designate individual GTV and respective PTV planning for each lesion. GTV will be all gross tumor identified by physical exam, additional clinical information and radiographic studies before induction chemotherapy. The GTV will be expanded by 3 to 5 mm to create PTV. PTV can be modified at the discretion of the treating physician for the constraints of normal tissue tolerance and to avoid extension beyond the skin.
- 4. **Field Size:** Appropriate field sizes will be determined at the time of simulation to treat gross disease and areas of potential microscopic disease. Field size and arrangement will be at the discretion of the attending radiation oncologist. The optimal field arrangement will be determined based on the treatment planning techniques employed. All fields must be treated during each treatment session. Only photon (x-ray) beams with photon energies 4-10 MV will be allowed. Because of uncertainties in beam commissioning resulting from electronic disequilibrium within small beam apertures, a minimum field dimension of 3.5 cm is required for any field used for treatment delivery. It is understood that this may exceed the technical requirements for small lesions (< 2.5 cm axial GTV dimension or < 1.5 cm craniocaudal GTV dimension). In such cases, the prescription dose is still prescribed to the edge of the defined PTV. This minimum field dimension does not apply to centers using tomotherapy or multiple pencil beam delivery systems.
- 5. **Treatment technique:** Blocking will be individualized for each patient. Either custom Cerrobend blocks, multileaf collimator or stereotactic cones will be acceptable.

**IMRT/VMAT**: IMRT/VMAT planning is preferred for SABR. IMRT/VMAT planning will depend on the planning system employed. We anticipate the optimal plan will use 7 to 11 gantry positions. Acceptable plans will encompass the PTV with the 95% isodose line. No more than 1% of the PTV should receive less than 95% of the prescribed dose. Plans should be reviewed to ensure that any part of the PTV getting less than 93% of the prescribed dose is at the edge of the volume. In no case should a central area of the PTV receive less than 95% of the prescribed dose. No more than 20% of the PTV should receive more than 110% of the prescribed dose.

3D Conformal Radiotherapy: Three-dimensional coplanar or non-coplanar beam arrangements will be custom designed for each case to deliver highly conformal prescription dose distributions. Non-opposing, non-coplanar beams are preferable. Typically,  $\geq 10$  beams of radiation will be used with roughly equal weighting. Generally, more beams are used for larger lesion sizes. When static beams are used, a minimum of seven non-opposing beams should be used. For arc rotation techniques, approximate rotation of 340 degrees (cumulative for all beams) should be utilized. For this protocol, the isocenter is defined as the common point of gantry and couch rotation for the treatment unit. Field aperture size and shape should correspond nearly identically to the projection of the PTV along a beam's eye view (i.e., no additional "margin" for dose buildup at the edges of the blocks or MLC jaws beyond the PTV). The only exception will be when observing the minimum field dimension of 3.5 cm when treating small lesions (see above). As such, prescription lines covering the PTV will typically be the 60-90% line (rather than 95-100%); however, higher isodoses (hotspots) must be manipulated to occur within the target and not in adjacent normal tissue. The plan should be normalized to a defined point corresponding closely to the center of mass of the PTV. For 3D techniques, acceptable plans will encompass the PTV within the 95% isodose line. The dose variation in the PTV will be +20% and -5% of the prescription point dose.

**Dose Fractionation:** Isodose calculations in the axial, sagittal, or coronal planes are required. In addition, dose volume histograms for the GTV and the spinal cord are required.

**SBRT** Radiation will be delivered in 800 to 880 cGy fractions to a total dose of 4000 to 4400 cGy (5 fractions total). Tumors <25 cm³ should receive 800 cGy per fraction for 5 fractions to 40 Gy; tumors ≥25 cm³ should receive 880 cGy per fractions for 5 fractions to 44 Gy. Each fraction will be given > 40 hours from the prior fraction (i.e. at least every other day) over a 2.5 week period. Ideally, treatment should be completed within 10 days. However, in case of holidays or unforeseen circumstances, treatment can be completed within 2.5 weeks.

The dose per fraction is to be prescribed to the prescription line at the edge of the PTV.

**Normal Tissue Constraints/Dose Volume Histograms:** The dose limit to the spinal cord will vary depending upon the technique used. All attempts should be made to limit the spinal cord dose to < 1000 cGy. The **cumulative** spinal cord dose should not exceed 5000 cGy at the equivalent dose of 2 Gy per fraction (EQD2) for all patients. In cases where cumulative spinal cord doses exceeds 5000 cGy, the **cumulative** maximum spinal cord dose may be as high as 5500 cGy at the equivalent dose of 2 Gy per fraction (EQD2) ONLY for patients where the interval between initial radiotherapy and re-irradiation is  $\geq$  2 years. The **cumulative** brainstem dose should not exceed 6000 cGy at the equivalent dose of 2 Gy per fraction (EQD2) for all patients. If prior radiotherapy plans are not available to assess the cumulative spinal cord dose, then the spinal cord dose from the initial radiotherapy plan should be assumed to be 5000 cGy. Equivalent doses will be estimated using the equation: Equivalent dose in 2Gy fractions (EQD2) = D x ({d + ( $\alpha/\beta$ )}/{2 + ( $\alpha/\beta$ )}). The  $\alpha/\beta$  ratio will be assumed to be 1 for the cervical spinal cord and 2 for the brainstem. Isodose calculations in the axial, sagittal, or coronal planes are required. In addition, dose volume

histograms for the planning treatment volumes and the following OARs are brachial plexus, carotid artery, parotid, cochlea, optic nerves, optic chiasm, larynx, esophagus. No more than 5% of any OAR or any other normal tissue should receive doses in excess of 110% of the primary PTV dose. Ultimate inclusion of the normal structures and exceptions from the above guidelines will be made at the discretion of theattending Radiation Oncologist.

The radiotherapy safety monitoring committee (RSMC): All radiation plans and dose statistics/dose volume histograms will be reviewed prior to initiating treatment by the RSMC. The RSMC is an independent safety monitoring committee formed by several radiation oncologists with expertise in the SBRT techniques and not involved in the study.

# Supportive Guidelines

- Antiemetics will be ordered at the discretion of the attending physician.
- Use of a feeding device is recommended for high-risk patients. Placement of a feeding device is left to the discretion of the treating physician/investigator. Commonly applied criteria for feeding device placement include
  - i. Loss of > 10% of body weight from the start of therapy
  - ii. Dehydration or inability to maintain adequate oral hydration
  - iii. Inability to maintain intake of > 25 kcal/kg of ideal body weight
- During radiotherapy patients may receive instructions for oral hygiene and prescriptions to include:
  - i. Oral nystatin or fluconazole (100mg QD)
  - ii. Viscous lidocaine HCl (Xylocaine®) solution) and/or Grade I mouthwash 10ml QID, swish and spit

Table 5: Grade I mouthwash (Magic Mouthwash)

| Lidocaine, Viscous (2%) | 50 mL |
|---------------------------------------|--------|
| Diphenhydramine elixir (12.5 mg/5 mL) | 50 mL |
| Sodium bicarbonate injection | 100 mL |
| Normal saline irrigation | 500 mL |
| Total volume | 700 mL |

- iii. Normal saline mouthwash 10ml QID swish and spit
- iv. Natural Care Gel (or similar product) BID during chemoradiotherapy and TID during rest week.
- v. Vigilon (or similar product) to be applied to open wounds during chemoradiotherapy.

- vi. Silvadene cream to open wounds followed by zinc oxide cream and then Telfa dressings BID during rest week (N.B.: discontinue Silvadene and zinc oxide creams 1 day prior to radiotherapy).
- vii. Aquaphor (or similar brand) cream to lips PRN.
- viii. Adequate analgesia is essential to maintain oral intake and patient comfort. Narcotic analgesics are usually necessary and should be used at the physician/investigator discretion.
  - ix. Therabite for trismus if appropriate.
  - x. Replacement for electrolyte imbalances when applicable.
- Prior to discharge of the patients after a cycle of chemoradiation, a CBC and platelet count, and determination of serum electrolytes, including creatinine will be done
- Use of intravenous home hydration is strongly recommended in patients with inadequate oral intake: normal saline 1000ml IV QD during rest week (days 6-14).
- If Hgb < 10, patients should generally be transfused an amount sufficient to increase Hgb to ≥ 10. The Hgb level should be maintained > 11 mg/dl for the duration of chemoradiotherapy in all patients.

#### 8 STUDY PROCEDURES

Study procedures should be completed as outlined in the Schedule of Events. Section 6.1 summarizes the trial procedures to be performed at each visit. Individual trial procedures are described in detail below.

**8.1** Schedule of Events (SoE)
Any treatment delays for less than five days will not be considered a study deviation.

| | Screenir | ng Phase | | | | | | | | | Treati | ment P | hase | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment Encounter | Part 1 | Part 2 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 |
| Scheduling Window | (-28 to<br>1) | (-14 to<br>-1) | Day<br>1 | Day<br>8 | Day<br>15 | Day<br>18 | Day<br>22 | Day<br>25 | Day<br>29 | Day<br>31 | Day<br>52 | Day<br>73 | Day<br>94 | Day<br>115 | Day<br>136 | Day<br>157 | Day<br>178 | Week 26<br>onwards <sup>g</sup> | End of<br>Study <sup>h</sup> |
| Informed Consent | X | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion<br>Criteria | X | | | | | | | | | | | | | | | | | | |
| Demographics and<br>Medical History | Х | | | | | | | | | | | | | | | | | | |
| Concomitant<br>Medication Review <sup>e</sup> | Х | | Х | Х | Х | | | Х | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Physical Examination <sup>e</sup> | | X | X | Х | X | | | X | | X | Х | X | Х | Х | X | Х | X | Хg | Х |
| Vital Signs and Weight <sup>e</sup> | | X | X | | X | | | | | X | | X | | Х | | Х | | Хg | Х |
| ECOG Performance <sup>e</sup><br>Status | | Х | Х | | Х | | | | | X | | Х | | Х | | Х | | Χg | Х |
| Pregnancy Test- Urine or Serum β-HCG | | Х | | | | | | | | | | | | | | | | | |
| PT/INR AND aPTT | | Х | | | | | | Χ | | Х | Χ | Х | X | Х | Х | Х | Х | Х | |
| CBC & Serum<br>Chemistry <sup>a</sup> | | X | Χ <sup>I</sup> | X | Х | | | X | | X | Х | X | Х | Х | X | Х | X | Xg | Х |
| Urinalysis | | Х | | | | | | | | | | Х | | Х | | Х | | $\mathbf{X}^{f}$ | Х |
| T3, FT4 and TSH | | Х | | | | | | | | | | | Х | | | | | Χ <sup>f</sup> | х |
| ECG | | Χ <sup>i</sup> | | | | | | | | | | | As clini | cally ne | eded | | | | |
| Tumor Imaging - CT Preferred <sup>b</sup> | X | | | | | | | | | | X | | | X | | | X | Xp | Х |
| Tissue Biopsy <sup>j</sup> | Х | | $\mathbf{X}^{\mathbf{k}}$ | Χ | | Х | | | | | | | X <sup>m</sup> | | | | | | |
| Correlative Blood Collection <sup>c</sup> | | Х | | Х | | Х | Х | | | | | | Xc | | | | | | Хc |
| SBRT | | | | | Х | Х | Χ | Χ | X | | | | | | | | | | |
| OBP-301 <sup>d</sup> | | | Х | X | | X | | Х | | Х | Х | Х | X | X | X | X | Х | Χ | |
| Pembrolizumab<br>Administration <sup>d</sup> | | | | Х | | | | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | |
| Review Adverse Events | | | X | Х | X | | | X | | X | Х | X | Х | Х | X | Х | X | Хg | Х |

- a. Serum chemistry includes sodium, potassium, chloride, bicarbonate, blood urea nitrogen, creatinine, glucose, AST, ALT, Alk Phos, lactate dehydrogenase, bilirubin (total and direct), total protein, albumin, calcium, magnesium and phosphorous.
- b. Tumor imaging studies preferably CT scans of chest/abdomen/pelvis should be performed every three cycles of pembrolizumab after week 26 until end of study.
- c. Correlative blood collection will be done during screening phase (-14 to -1), on day 1 (prior to drug administration), day 8, day 18, day 22, day 94 (optional), and at the end of study. Baseline correlative bloods can be collected on study Day 1 if missed during screening. Correlative blood draws will be done pre-dose if treatment is given on the same day.
- d. Pembrolizumab and OBP-301 can be administered with a  $\pm$  5 day window in accordance with the above treatment plan. Pembrolizumab will be administered on day 8 and then every 3 weeks  $\pm$  5 days starting on day 31.
- e. Baseline assessment should be performed within 5 days of administrating first dose of OBP-301.
- f. Urinalysis, T3, FT4 and TSH should be performed every 3rd cycle of pembrolizumab thereafter until end of study.
- g. From week 26 and onwards, concomitant medication review, physical exam, vitals/weight, ECOG performance status, CBC, comprehensive serum chemistry and review of adverse events should be performed every 3 weeks until end of study.
- h. End of study will occur 28 days (+/- 5 days) following study removal, disease progression, or following 1 year on treatment. Patients may still be followed for survival for up to 96 weeks from study start.
- i. 12-lead ECG will be recorded after the patient has rested for 5 minutes
- j. Tumor biopsy may be needed during screening phase for PD-L1 testing if there is no archival tissue available. If there is no archival tissue available, tissue collection for PD-L1 testing and correlative studies will be performed during screening phase. If patient is determined to be PD-L1 testing and correlative studies will be performed during screening phase.
- L1 negative they are not eligible for the study and the additional tissue that was collected for correlative studies will be returned to pathology.
- k. If biopsy was performed during screening phase to confirm PD-L1 status, No biopsy should be performed on Day 1. Day 1 biopsy only to be performed for correlative studies if a biopsy was not performed at baseline.
- 1. Only needed, if screening CBC and chemistry done more than 7 days prior to first cycle of pembrolizumab.
- m. An optional biopsy will be done on Day 94 +/- 5 days.

# 8.1.1 Screening Visit

- Informed consent
- Demographics
- Medical history
- Concomitant Medications
- Physical exam
- Vital signs and weight
- ECOG performance status (Appendix A: ECOG Performance Status Criteria)
- Urine or Serum Pregnancy Test
- PT/INR and aPTT
- Complete Blood Count (CBC) with differential
- Serum chemistry
- Urinalysis
- T3, FT4 and TSH
- ECG
- Tumor Imaging CT preferred
- Tumor Biopsy/Archival biopsy (for PD-L1 status)
- Correlative Blood Collection

# 8.1.2 Treatment Phase

Pembrolizumab infusions will be administered on day 8 and then every 3 weeks  $\pm$  5 days starting on day 31 until disease progression or patient is withdrawn for another reason or up to one year if no progression.

OBP-301 only, is to be administered on D1, then in combination with pembrolizumab on D8, then in combination with SBRT on D18 and D25, then again in combination with pembrolizumab every 3 weeks on days D31, D52, D73, D94, D115, D136, D157 and D178. On days that both Pembrolizumab and OBP-301 are administered, there is no specificity to which drug should be administered first. The target tumor will be injected with OBP-301 up to 12 times during the entire study.

All patients will receive OBP-301 at a concentration of  $1x10^{12}$  viral particles/ml injection. Volume to be injected is up to 4ml and will depend on lesion size i.e. the longest diameter of the lesion) (see Table 1, section 5.2.2 above).

### 8.1.3 Follow up Phase

Patients with disease progression will be followed every 3 months for survival for up to 2 years after last treatment. If patient unable to come for follow up, the assessment can occur by telephone or some other remote monitoring.

# 8.1.4 Patient Withdrawal Criteria

In accordance with applicable regulations, a participant has the right to withdraw from the study, at any time and for any reason, without prejudice to his future medical care.

Withdrawal from the study and therapeutic measures taken shall be at the discretion of the Investigator. A full explanation for the discontinuation from the study should be made in the participant's medical records and in the eCRF.

Premature discontinuation from active study participation may occur at any time due to any of the following reasons:

- Any situation where, in the opinion of the Investigator or the Medical Monitor, continued participation in the study would not be in the best interest of the patient.
- Positive pregnancy test
- Patient initiates other anti-cancer therapy. The anti-cancer therapy will be documented in the medical record and eCRF.
- Progressive neoplastic disease, unless the Investigator feels this may be pseudoprogression, in which case the patient may remain on study until the next evaluation for extent of disease.
- An intercurrent illness or AE that requires concomitant medication that precludes further study participation
- Patient is unable or unwilling to comply with study procedures.
- Patient is lost to follow-up.
- Patient withdraws consent.
- Termination of the study by the Sponsor.
- Request by a Health Authority.

In addition, the Sponsor will discontinue a patient from active study treatment for any of the following criteria (subjects will continue to be followed as apprioprate for outcomes and toxicities:

- Patients who experience a Grade 4 hematologic toxicity or a Grade 3 or greater non-hematologic toxicity attributable to OBP-301 or that has not resolved to Grade 1 (or basline) within 2 weeks of onset.
- OBP-301 injection will be delayed for any ongoing Grade 2 toxicity at the time of the next scheduled injection after consultation with the Principal Investigator. Patients who require a delay of OBP-301 injection of > 4 weeks (i.e., approximately 6 weeks from the previous injection) due to lack of resolution to Grade 1 toxicity will be discontinued from the study after consultation with Medical Monitor and Principal Investigator.

Psuedo-progression occurs very rarely in head and neck cancer. If the patient is asymptomatic, after apparent disease progression (PD) is observed as per iRECIST, a biopsy of the lesion should be done to evaluate response. If progression is documented by the biopsy, administration of OPBP-301 will be discontinued. If response is confirmed by the biopsy, administration of OBP-301 may be continued. Immune-related disease progression (irPD) will be confirmed if the increase in tumor burden is  $\geq 25\%$  relative to nadir (minimum recorded tumor burden). The confirmation is completed by a repeat, consecutive assessment no less than 4 weeks from the date the disease progression was first documented. If in the opinion of the investigator, at the repeated scan, the disease progression is not clinically significant, then the patient may continue to receive OBP-301 treatment

The reason(s) for premature study discontinuation/withdrawal will be documented along with the date of withdrawal. AEs should be documented according to the study calendar.

For all patients who discontinue, a Final Visit will be performed within  $28 \pm 5$  days after the last IP administration (see study calendar). If a participant is withdrawn because of an AE, the Investigator must arrange for the participant to have appropriate follow-up care until the AE is resolved or has stabilized. Unresolved AEs will be followed until the last scheduled follow-up visit or until the Investigator and Medical Monitor determine that further follow-up is no longer indicated. Investigators should attempt to collect the survival information as dictated by the Schedule of Events in the Study calendar.

Patients who discontinue the active study participation will not be replaced.

Any enrolled patients who are discontinued before study dosing will be documented as screen failures in the eCRF and replaced. No follow-up is required for these patients.

# 8.2 Informed Consent Form (see appendix)

Each patient is required to provide informed consent before participating in the study.

Before performance of any study procedures, potential patients will attend a screening session at which time they will be provided with full information concerning details of the study assessments and procedures. They will also be provided with the ICF. Before being asked to sign the ICF, patients will be given time to review the study information and ask any questions. A copy of the signed ICF must be provided to the patient.

# 8.3 Demographic Data and Baseline Characteristics

Gender, date of birth, height, and weight, as well as race and ethnic origin will be recorded for each patient and age and body mass index calculated from these data.

# 8.4 Medical History, Concomitant Disease, Previous and Ongoing Medications

A detailed medical history, including surgical and cancer history, will be recorded and will include any conditions reported by the patient or noted by the Investigator in each body system. Medical history is defined as any condition that started and ended before the Screening Visit. A concomitant disease is defined as any condition detected at the Screening Visit that started after ICF signature or was started before the Screening Visit and is still ongoing at the Screening Visit.

Prior medication taken before the Screening Visit and any concomitant medication will be documented. Prior medication is defined as any medication taken within 4 weeks of screening visit. Concomitant medications are those medications which the patient is currently taking at any particular visit.

Records should include the drug name (preferably both generic and trade name), route of administration (e.g., oral, intravenous), injection and frequency (expressed in metric units, for example, mg, mL, or IU), indication, and the start and, if applicable, the stop date (day, month,

and year). Therapy changes (including changes of regimen) during the study have to be documented. All concomitant medications will be recorded in the eCRF.

# 8.5 Safety Assessments

#### **8.5.1** Adverse Events

Definitions, management of, and special considerations for AEs are provided in Section 7. Adverse events will be collected at each contact with the patient. Questions regarding the presence of adverse events should be open-ended without leading the patient.

# 8.5.2 Physical Examination

The physical examination is to be conducted by the Investigator or designated fully trained representative. Performance status will also be determined at screening as well as at each subsequent visit as oulined in the section study schedule. Patients will be graded according to the ECOG Performance Status Scale.

| Performance<br>Status | Definition |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction. |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work. |
| 2 | Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours. |
| 3 | Capable of limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | Completely disabled; cannot carry on any self-care; totally confined to bed or chair. |

# 8.5.3 Vital Signs

Vital signs will include measurements of heart rate, systolic and diastolic blood pressures while the patient is in a seated position, and temperature.

#### 8.5.4 Electrocardiogram

During screening of patients, a standard baseline 12-lead ECG will be recorded after the patient has rested for 5 minutes. The Investigator or designee will review all ECGs. The following parameters will be documented: rhythm, heart rate, PR interval, QRS interval, QT interval, and QTc. Every ECG must be assessed as normal, abnormal – clinically not significant, or abnormal – clinically significant. A diagnosis must be provided in the eCRF for all ECGs assessed as

abnormal – clinically significant. If clinically indicated, additional ECGs may be obtained during the study.

# 8.5.5 Laboratory Assessments

# 8.5.5.1 Clinical Chemistry, Hematology, Coagulation Parameters, and Urine Analysis for Safety Panel

Following table illustrates laboratory assessments, which will be performed at prescribed intervals as per schedule of events.

 Table 4
 Clinical Laboratory Parameters for Safety Panel

| Hematology | Coagulation | Serum Chemistry | <b>Urine Analysis</b> |
|---|---|---|---|
| <ul> <li>Hemoglobin</li> <li>Hematocrit</li> <li>Red blood cell count</li> <li>White blood cell (WBC) count</li> <li>Platelet count</li> <li>WBC differentials</li> </ul> | <ul> <li>International normalized ratio</li> <li>Prothrombin time</li> </ul> | <ul> <li>Sodium</li> <li>Potassium</li> <li>Chloride</li> <li>Bicarbonate</li> <li>Blood urea nitrogen</li> <li>Creatinine</li> <li>Glucose</li> <li>Alanine transaminase</li> <li>Aspartate transaminase</li> <li>Alkaline phosphatase</li> <li>Lactate dehydrogenase</li> <li>Bilirubin (total and direct)</li> <li>Total protein</li> <li>Albumin</li> <li>Calcium</li> <li>Magnesium</li> <li>Phosphorous</li> </ul> | <ul> <li>pH</li> <li>Specific gravity</li> <li>Glucose</li> <li>Ketones</li> <li>Bilirubin</li> <li>Hemoglobin</li> <li>Protein</li> <li>Microsopic if any dipstick value 2+ or greater</li> </ul> |

# 8.5.5.2 Pregnancy Testing and Post-Menopausal Status

A serum or urine pregnancy test will be performed on all women of childbearing potential at Screening.

The post-menopause is defined as the time after which a woman has experienced 12 consecutive months of amenorrhea (lack of menstruation) without a period. If a woman

claims she is post-menopausal, but has had her menses within 12 months, a follicle stimulating hormone (FSH) test must be performed and must be within acceptable limits of the post-menopausal status. If the post-menopausal status of a female is confirmed, the pregnancy tests will not be performed.

All pregnancies detected during the study must be reported and handled as described in Section 7.2.

# **8.6** Efficacy Assessments

# **8.6.1** Imaging Assessment for the Study

All the patients who enrolled into study will undergo efficacy assessments for overall response rate, disease control rate, progression free survival and overall survival, as defined in Section 8.5. A baseline imaging study preferably CT scan of chest/abdomen/pelvis with IV contrast (permitting no contraindication to contrast) will be performed followed by CT scans at regular intervals at the treating physician discretion. The first CT scan will be performed at 9 weeks after the initial CT scan. While the patient is on study CT scans should be performed every 9 weeks (-1 week/+3 week window). Efficacy end points will be assessed according to RECIST 1.1 and iRECIST criteria.

#### 8.6.2 Definitions of Measurable and Non-Measurable Disease

#### **8.6.2.1** Measurable Disease

Tumor lesions: Must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of 10 mm by CT scan (CT scan slice thickness no greater than 5 mm).

Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be 15 mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.

# 8.6.2.2 Non-Measurable Disease

All other lesions, including small lesions (longest diameter <10 mm or pathological lymph nodes with 10 to <15 mm short axis) as well as truly non-measurable lesions. Lesions considered truly non-measurable include: leptomeningeal disease, ascites, pleural or pericardial effusion, inflammatory breast disease, lymphangitic involvement of skin or lung, abdominal masses/abdominal organomegaly identified by physical exam that is not measurable by reproducible imaging techniques.

# 8.6.3 Response Criteria

All patients will undergo re-evaluation imaging scans every nine weeks from the start of treatment as per the study schedule to determine response to treatment. Intervals between scans should not exceed 12 weeks. Following designations will be assigned according to RECIST 1.1 and iRECIST (see appendix below for differences in RECIST 1.1 and iRECIST). The

primary end point-response criteria is RECIST 1.1 in both injected and uninjected target lesions. iRECIST is only a secondary end point response criteria.

# 8.6.3.1 Complete Response (iCR)\*

Defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

# 8.6.3.2 Partial Response (iPR)\*

At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

# 8.6.3.3 Progressive Disease (PD)\*

At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.

Unconfirmed PD (iUPD) requires confirmation, which is done on the basis of observing either a further increase in size (or in the number of new lesions) in the lesion category in which progression was first identified in (i.e., target or non-target disease), or progression (defined by RECIST 1.1) in lesion categories that had not previously met RECIST 1.1 progression criteria. However, if progression is not confirmed, but instead tumor shrinkage occurs (compared with baseline), which meets the criteria of iCR, iPR, or iSD, then the bar is reset so that iUPD needs to occur again (compared with nadir values) and then be confirmed (by further growth) at the next assessment for confirmed progressive disease (iCPD) to be assigned. If no change in tumor size or extent from iUPD occurs, then the timepoint response would again be iUPD.

# 8.6.3.4 Stable Disease (iSD)\*

Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

\* May have had unconfirmed progressive disease (iUPD) (1 or more instances), but not confirmed progressive disease (iCPD), prior to complete response (iCR), partial response (iPR) or stable disease (iSD). "i" indicates immune responses assigned using iRECIST.

# 8.6.4 Determination of Tumor Stage According to Tumor, Lymph Nodes, Metastasis (TNM) Classification

In some circumstances, it may be difficult to distinguish residual disease from normal tissue. When the evaluation of CR depends on this assessment, it is recommended that the residual lesion be investigated (fine needle aspirate/biopsy) before confirming the complete response status.

# 8.7 Biopsies and Immune Monitoring (optional)

In order to observe a potential response in the non-injected lesions, if several tumors are present, biopsies will be taken at baseline (Day 1) and on Day 18 both from an injected tumor and a non-injected tumor and a comparison will be done between them.

Standard fine needle biopsies will be taken on the following days:

- 1. Day 1, prior to therapy,
- 2. Day 8, prior to therapy (to see the effect of OBP-301 alone),
- 3. Day 18, prior to therapy (to see the effect of OBP-301 together with pembrolizumab). Given the fact that three biopsies will be done within approximately 3 weeks, special attention will be given to potential side effects (i.e. bleeding, etc.) that can be associated with the biopsy procedures.
- 4. Optional on Day 94 +/- 5 days (to see the effect of OBP-301 + pembrolizumab + SBRT).

Correlative blood samples will be taken before the start of study treatment, during treatment and post-treatment as described in the section of study schedule. Blood and biopsy samples will be retained for future research if informed consent has been obtained from the patient.

#### 9 ADVERSE EVENTS

#### 9.1 Definitions

# 9.1.1 Definition of an Adverse Event

An AE is any event, side effect, or other untoward medical occurrence that occurs in conjunction with the use of a medicinal product in humans, whether or not considered to have a causal relationship to this treatment. An AE can, therefore, be any unfavorable and unintended sign (that could include a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

Events meeting the definition of an AE include:

- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after IP administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either IP or a concomitant medication (overdose per se will not be reported as an AE/SAE).

"Lack of efficacy" or "failure of expected pharmacological action" per se will not be reported as an AE or SAE. However, the signs and symptoms and/or clinical sequelae resulting from lack of efficacy will be reported if they fulfil the definition of an AE or SAE.

Events that do not meet the definition of an AE include:
- Medical or surgical procedure (e.g., appendectomy). The condition that leads to the procedure is an AE.
- Situations where an untoward medical occurrence did not occur (e.g., social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

If there is evidence of an AE through report or observation, the Investigator or designee will evaluate further and record the following information:

- Date of onset and resolution
- Classification of 'serious' or 'non-serious'
- Severity
- Causality/relation to study treatment
- Action taken regarding IP (no action taken, study treatment interrupted, study treatment discontinued)
- Medication or additional treatment (no medication additional treatment, concomitant medication, non-drug therapy, other)
- Outcome /Status (recovered, recovered with sequelae, recovering, ongoing, fatal unknown)

# 9.1.2 Severity of an Adverse Event

The intensity of AEs/SAEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 (dated 27 Nov 2017) <sup>65</sup>.

Should an event be missing in the NCI-CTCAE, the following 5-point scale is to be used:

- Mild: Discomfort noticed, but no disruption of normal daily activity
- Moderate: Discomfort sufficient to affect normal daily activity
- Severe: Inability to work or perform normal daily activity
- Life-threatening: Risk of death at the time of the event
- Fatal: The patient died

The correspondence between the 2 scales is as follows:

| NCI-CTCAE | 5 point scale |
|-----------|------------------|
| 1 | Mild |
| 2 | Moderate |
| 3 | Severe |
| 4 | Life-threatening |
| 5 | Fatal/Death |

NCI-CTCAE = National Cancer Institute Common Terminology Criteria for Adverse Events

#### 9.1.3 Causal Relationship of an Adverse Event

Causal relationship of an adverse event to the IP will be assessed by the Investigator as follows:

Not related: The event is clearly related to other factors such as the participant's clinical state, therapeutic interventions or concomitant drugs

administered to the participant. This is especially so when an event

occurs before the commencement of treatment with the IPs.

Unlikely: The experience was most likely produced by other factors such as the

participant's clinical state, therapeutic interventions or a concomitant drug administered to the participant and does not follow a known

response to the trial IP.

Possible: The experience follows a reasonable temporal sequence from the time

of IP administration and/or follows a known response to the trial IP, but could have been produced by other factors such as the participant's clinical state or other therapeutic interventions or concomitant drugs

administered to the participant.

Probable: The experience follows a reasonable temporal sequence from the time

of IP administration and follows a known response to the trial IP, and cannot be reasonably explained by other factors such as the participant's clinical state or other therapeutic interventions, or concomitant drugs

administered to the participant.

Definite: The experience follows a reasonable temporal sequence from the time

of IP administration and follows a known response to the trial IP, and cannot be reasonably explained by other factors such as the participant's clinical state or other therapeutic interventions or concomitant drugs administered to the patient and in addition one or more of the following:

Occurs immediately following trial IP administration

o Improves on stopping the trial IP

Reappears on repeat exposure

#### 9.1.4 Definition of a Serious Adverse Event

An SAE is any untoward medical occurrence regardless of the grade that:

- results in death,
- is life-threatening,
- requires inpatient hospitalization or prolongation of existing hospitalization,
- results in persistent or significant disability/incapacity, or,
- is a congenital anomaly/birth defect.

Important medical events that may not be one of the above may be considered an SAE by the Investigator when, based upon appropriate medical judgement, are considered clinically significant and may jeopardize the participant, or may require medical or surgical intervention to prevent one of the outcomes listed above.

"Life-threatening" means that the participant was at immediate risk of death from the experience that, had it occurred in a more serious form might have caused death.

A congenital anomaly in an infant born to a mother who was exposed to the IP during pregnancy is considered an SAE. Procedures for notification of pregnancies and follow-up are described in Section.

# 9.1.5 Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events and Serious Adverse Events

Abnormal laboratory findings (e.g., clinical chemistry, hematology, and urinalysis) or other abnormal assessments (e.g., ECG, X-rays, and vital signs) per se are not reported as AEs. However, those abnormal findings that are deemed **clinically significant** or are associated with signs and/or symptoms must be recorded as AEs if they meet the definition of an AE (and recorded as an SAE if they meet the criteria of being serious) as described previously. Clinically significant abnormal laboratory or other abnormal findings that are detected after consent or that are present at the time of consent and worsen after consent are included as AEs (and SAEs if serious).

The Investigator should exercise his or her medical and scientific judgment in deciding whether an abnormal laboratory finding or other abnormal assessment is clinically significant. Usually, the abnormality should be associated with a clinically evident sign or symptom, or be likely to result in an evident sign or symptom in the near term, to be considered clinically significant. A clinically significant laboratory abnormality in the absence of clinical symptoms may jeopardize the participant and may require intervention to prevent immediate consequences. For example, a markedly low serum glucose concentration may not be accompanied by coma or convulsions, yet be of a magnitude to require glucose administration to prevent such sequelae.

#### 9.2 Documenting Adverse Events

Any AE occurrence (spontaneously volunteered and enquired for, as well as observed AEs) during the study must be documented in the patient's medical records in accordance with the Investigator's normal clinical practice and on the AE page of the eCRF. SAEs that occur during the study must be documented in the patient's medical record, on the AE eCRF, and on the SAE form.

The Investigator should attempt to establish a diagnosis of the event based on the signs, symptoms, and/or other clinical information. In such cases, the diagnosis should be documented as the AE (and SAE if serious) and not the individual signs/symptoms.

If a clinically significant abnormal laboratory finding or other abnormal assessment meets the definition of an AE, then the AE eCRF page in the REDCap database must be completed as appropriate. In addition, if the abnormal assessment meets the criteria for being serious, the SAE form must also be completed. A diagnosis, if known, or clinical signs or symptoms if the diagnosis is unknown, rather than the clinically significant laboratory finding or abnormal assessment, should be used to complete the AE/SAE page. If no diagnosis is known and clinical signs or symptoms are not present, then the abnormal finding should be recorded. If an SAE report is completed, pertinent laboratory data should be recorded on the SAE form, with baseline values and copies of laboratory reports.

The SAE page should be completed as thoroughly as possible and signed by the Investigator before transmittal to Oncolys BioPharma Inc at safety@oncolys.com.

It is very important that the Investigator provide an assessment of the causal relationship between the event and the IP at the time of the initial report, as this will be useful for submissions to regulatory authorities.

# 9.2.1 Recording of Adverse Events

All adverse events will be recorded on a patient specific AE log after W1D1 and entered onto REDCap. The AE log will be maintained by the research staff and kept in the patient's research chart.

# 9.2.2 Reporting of AE to WCMC IRB

All adverse events will be recorded on a patient specific AE log after Day 1. The AE log will be maintained by the research staff and kept in the patient's research chart.

#### 9.2.3 Follow-up of Adverse Events and Serious Adverse Events

In this study, non-serious AEs will be reported in all participants from Treatment 1. Non-serious AEs reported from the time of consent to injecting on Day 1 will be recorded as medical history. Serious adverse events (SAEs) will be reported in all patients (enrolled and not enrolled) from the time of consent. Study procedure-related AEs will be evaluated specifically from the time of consent until the administration of OBP-301. Treatment-emergent AEs will be evaluated from the time of injecting with IP until the Final Visit. The Investigator is responsible to ensure that follow-up includes any supplemental investigations as may be indicated to elucidate as completely as practical the nature and/or causality of the AE/SAE. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.

All non-serious AEs that are ongoing at the Final Visit will be marked as ongoing on the AE eCRF page in the REDCap database.

All SAEs that are ongoing at the Final Visit must be followed until resolution, until the condition stabilizes, until the event is, in the opinion of the Investigator, stabilized or determined to be chronic, or until the participant dies or is lost to follow-up. SAEs that occur after the Final Visit, that are thought to be related to the administration of OBP-301, should be reported to Oncolys BioPharma Inc. or designee.

If a participant is withdrawn because of an AE, the Investigator must arrange for the participant to have appropriate follow-up care until the AE is resolved or has stabilized. Unresolved AEs will be followed until the last scheduled follow-up visit or until the Investigator and Medical Monitor determine that further follow-up is no longer indicated. Oncolys BioPharma Inc. may request that the Investigator perform or arrange for the conduct of supplemental measurements and/or evaluations. If a participant dies during participation in the study or during a recognized Follow-up Period, Oncolys BioPharma Inc. should be provided with a copy of any post-mortem findings, including histopathology.

# 9.2.4 Reporting of SAE to IRB

All SAEs occurring after study treatment on this study will be reported to the IRB according to the IRB policy, which can be accessed via the following link: http://researchintegrity.weill.cornell.edu/forms\_and\_policies/forms/Immediate\_Reporting\_Policy.pdf.

For WCM investigator-initiated studies, the following reporting guidelines apply:

a. A Mandatory MedWatch Form 3500A must be completed and sent to the FDA. Specific instructions on how to complete the MedWatch Form 3500A can be found on the FDA website.

b. If the protocol requires SAEs to be reported to an outside agency (i.e., to the supplier of the study drug), specific instructions will be stated in the protocol.

- c. If the study utilizes the WCM Data and Safety Monitoring Board (DSMB), a narrative of the event will be submitted to the Regulatory Coordinator on a modified SAE cover sheet. The completed form serves as acknowledgement of the SAE's occurrence and will be used to complete the DSMB periodic report. A copy should be filed in the regulatory binder.
- d. For multicenter studies, the multicenter core within the Quality Assurance Unit (QAU) will distribute the IND Safety Report

#### 9.2.5 Notification of Serious Adverse Event to Oncolys

An SAE must be reported by the Investigator within 24 hours of discovery if it occurs during the clinical study or within 28 days of receiving the IP, whether or not the SAE is considered to be related to the IP. An SAE report consists of the SAE form, the AE form, and the concomitant medication form. A copy of these forms must be e-mailed to the attention within 24 hours of discovery:

### E-mail: safety@oncolys.com

The Investigator should not wait to receive additional information to document fully the event before notification of a SAE, though additional information may be requested. Where applicable, information from relevant laboratory results, hospital case records, and autopsy reports should be obtained.

Instances of death, congenital abnormality, or an event that is of such clinical concern as to influence the overall assessment of safety, if brought to the attention of the Investigator at any time after cessation of IP administration and linked by the Investigator to this study, should be reported to.

All SAEs must be reported to the investigational site's IEC/IRB by the Investigator in accordance with their regulations.

Investigator should report applicable adverse events to FDA per 21 CFR 312.32. The applicable form, such CIMOS or Medwatch that Investigator reported to FDA must also be provided to Oncolys BioPharma Inc (safety@oncolys.com) when SAE was considered OBP-301 related. In the case of unexpected fatal or life-threatening suspected adverse reaction, Investigator should provide the FDA report form to Oncolys no later than 3 days following Oncolys' initial receipt of the information. Additionally, in the case of other SAE must be reported to FDA within 15 days of learning of the adverse event, investigator should provide the FDA report form to Oncolys no later than 7 days following Oncolys' initial receipt of the information.

Reporting of any SAEs to applicable regulatory authorities will be the responsibility of Oncolys BioPharma Inc. in compliance with local regulations.

#### 9.2.6 Notification of Suspected Unexpected Adverse Reactions

An unexpected adverse reaction is any untoward and unintended response that is related to the administration of the IP at any concentration that is not consistent with the applicable version of the Investigator's Brochure [32].

All suspected unexpected serious adverse reactions (SUSARs) will be the subject of expedited reporting in accordance with local requirements. All Investigators should follow-up SUSARs until the event is resolved or until, in the opinion of the Investigator, the event is stabilized or determined to be chronic. Post study SAEs that are deemed to be related to IP that occur after the patient has completed the clinical study must be reported by the Investigator to Oncolys BioPharma Inc.

## 9.2.7 Notification of Pregnancies

All pregnancies in female patients and female partners of male patients receiving IP will be recorded from treatment until 90 days after the patient has completed therapy.

Should a patient or male patient's partner become pregnant or suspect she is pregnant while participating in this study, or in the 90 days following when the patient received the last injection of IP, the treating Investigator should be informed immediately. All pregnancies will be reported on a pregnancy report form and submitted to safety along the same timelines as an SAE.

The IEC/IRB and Oncolys BioPharma Inc. will be informed. The patient will be asked to provide information on the outcome of the pregnancy, including premature termination should the case arise. For pregnancies in a female partner of a male patient consent to follow-up on the pregnancy will be obtained in agreement with the US Health Insurance Portability and Accountability Act (HIPAA) and other local laws and regulations as outlined in Section. Pregnancy outcomes will be reported on a pregnancy follow-up report form.

Spontaneous miscarriage and congenital abnormalities will be reported as SAEs. The Follow-up Period for any and all pregnancies will be deemed to have ended when the health status of the child has been determined on its birth and followed up for 8 weeks after the birth for any potential abnormalities.

Full details will be recorded on the withdrawal page of the eCRF.

#### 9.3 Multicenter Study Monitoring

The study will be monitored by the Weill Cornell Multicenter Study group, according to the Clinical Trial Monitoring Plan, which addresses site qualification, regulatory documentation, and site monitoring and auditing.

#### 10 STATISTICAL ANALYSES

#### 10.1 General Considerations

The statistical evaluation will be performed using SAS®, version 9.4 or later.

All data will be presented in listings, ordered by patient, unless otherwise specified.

Descriptive statistics for continuous variables (number of patients [n], number of patients with missing data, mean, standard deviation, minimum and maximum) and categorical data (n, percent, number of patients with missing data, by category) will be presented.

#### 10.2 Definitions for Statistical Data Analysis

The following definitions were used in the assessments of safety and efficacy.

All patients who receive at least one injection of OBP-301 will be included in the Safety Population and are analysed according to the actual treatment received. Any patient that has at least one radiographic assessment for response will be included in the Efficacy Population.

#### 10.3 Handling of Missing Values and of Values outside the Detection Limits

Descriptive statistics for demographics, body weight, vital signs, and ECG data will be calculated from actual data only, with the number of actual data points used for the calculation of the summary statistics reported.

For censored safety lab data (i.e., hematology, clinical chemistry and urinalysis results that are outside the limit of quantification) the actual values reported by the laboratory (e.g., "< 2" for bilirubin) will be presented in the data listings. For the calculation of summary statistics, safety laboratory data values below the lower limit of quantification (LLOQ) will be set to ½ the LLOQ.

#### 10.3.1 Data Collection

The data collection plan for this study is to utilize REDCap to capture treatment, toxicity, efficacy, and adverse event data for all enrolled patients.

#### **10.3.2** REDCap

REDCap (Research Electronic Data Capture) is a free data management software system that is fully supported by the Weill Cornell Medical Center CTSC. It is a tool for the creation of customized, secure data management systems that include Web-based data-entry forms, reporting tools, and a full array of security features including user and group based privileges, authentication using institution LDAP system, with a full audit trail of data manipulation and export procedures. REDCap is maintained on CTSC-owned servers that are backed up nightly and support encrypted (SSL-based) connections. Nationally, the software is developed, enhanced and supported through a multi-institutional consortium led by the Vanderbilt University CTSA.

#### 10.4 Analysis Populations

#### **10.4.1 Safety Population**

All patients who receive at least one injection of OBP-301 will be included in the Safety Population and are analysed according to the actual treatment received.

## 10.4.2 Evaluable Population

Any patient that has at least one radiographic assessment on study for response will be included in the Efficacy Population. Imaging studies preferably CT scan of the chest/abdomen/pelvis will be performed every 9 weeks as per the study schedule. Patients will be evaluated according to RECIST v1.1 criteria. Definitions of response evaluation are detailed in section 6.6 for further explanation. Only those patients whose response can be measured according to RECIST v1.1 will be included in this population. Inevaluable patients will be replaced.

### 10.4.3 Intent-to-Treat (ITT) Population

All patients who are enrolled and allocated to treatment are included in the intent-to-treat population analysis.

# 10.4.4 Per-Protocol (PP) Population

Per-Protocol population will only include individuals who completed all twelve doses of OBP-301 and followed the study protocol.

#### 10.5 Efficacy Analysis

## 10.5.1 Primary Efficacy Endpoint

The primary efficacy endpoint will be the objective response rate (RR), as measured by RECIST 1.1 criteria.

Objective response rate is defined as the sum of partial responses (PR) plus complete responses (CR) as defined by RECIST v1.1 criteria.

# 10.5.2 Secondary Efficacy Endpoints

Secondary efficacy endpoints include the disease control rate (DCR), duration of response (DoR), progression-free survival (PFS), and overall survival (OS). A secondary efficacy endpoint will also be the objective response rate (ORR), as measured by RECIST 1.1 and iRECIST 1.1 criteria.

DOR is defined as the duration that subjects who have responded to combination therapy remain without disease progression.

DCR is defined as the percentage of patients who have achieved complete response, partial response and stable disease.

PFS is defined as time from registration to progression or death due to any cause. Progression is defined as radiologic progression of disease by RECIST v1.1 criteria.

OS is defined as the time from registration until death from any cause,

#### 10.5.3 Exploratory Analysis

Correlative endpoints include the following:

- To monitor viral replication post-treatment, viral protein expression in biopsies will be examined by immunostaining (Hexon) or FACS (CAR).
- To examine the tumor-immune microenvironment prior to and following OBP-301 and pembrolizumab therapy as assessed by immunohistochemistry.
- To examine and characterize the immune infiltrate by multi-parameter flow cytometry.
- To identify possible biomarkers (i.e. exosomes, ctDNA) for response and mechanism of resistance by longitudinal profiling of patients before and after immunotherapy + OBP-301 + SBRT.

# Methods for Analysis

Endpoints involving response rates will be analysed by tabulating the response rates along with 95% confidence interval and number of patients with data for each time point that the endpoint is collected. Waterfall plots for tumor response (CR, PR, and ORR) will be provided.

Endpoints involving time to event or time to response will be analysed using survival analysis, including Kaplan-Meier plots. Median survival time with 95% confidence interval, 25th-75th percentiles will be provided.

Exploratory subgroup analyses for tumor response will be defined in the statistical analysis plan (SAP).

#### 10.6 Correlative Studies

The purpose of our correlative studies is to identify potential associations between biomarkers and certain outcomes and not to for identifying predictive biomarkers. All patients undergoing treatment with OBP-301 will have tissue biopsies along with correlative blood samples. In order to observe a potential response in the non-injected lesions, if several tumors are present, biopsies will be taken both from an injected tumor and a non-injected tumor and a comparison will be done between them. Tissue biopsies will be performed at:

- -At screening (day -14 to -1)
- -Day 1 BEFORE administering the first dose,
- -then Day 8 to see the effect of OBP-301 alone,
- -then Day 18, to see the effect of OBP-301 together with pembrolizumab,
- -then at Day 94 to see the effect of OBP-301 + pembrolizumab + SBRT.

Correlative blood samples will be taken before the start of study treatment, during treatment and post-treatment as described in the section of study schedule. Correlative studies are focused on a detailed and comprehensive evaluation of the tumor immune microenvironment as it

relates to induction of the anti-tumor immune response. Specific procurement and shipping instructions will be provided to participating sites upon study activation. Our specific correlative studies include the following:

# A. To detect viral replication in the tumor environment. To examine the tumor-immune microenvironment prior to and following OBP-301 and pembrolizumab therapy

In order to detect viral replication in the tumors, post-treatment with OBP-301, biopsies will be immunostained for adenovirus proteins (Hexon AB1056; Millipore, Burlington, M) <sup>65</sup>. In patients that the presence of the virus is not detected we will perform Coxackie Adenovirus Receptor (CAR) expression analysis by FACS<sup>68</sup>.

Also, we will perform detailed cellular characterization of head and neck tumors and their microbial environment towards better understanding of the factors that shape the response to immunotherapies and mechanism of resistance. To address this, we propose to perform single cell expression analysis and microbiome profiling of tissue samples collected from patients with esophageal/gastric tumors.

We will correlate the response to the oncolytic virus with the presence/absence of the virus using a Fisher exact test.

We hypothesize that surveying the immune infiltration in the context of immunotherapy and OBP-301 will provide important biomarker for response to treatment. To address this, we propose the following analysis: Identify and quantify the cellular composition of tumor and adjacent normal tissues from head and neck cancer patients. In order to observe a potential response in the non-injected lesions, if several tumors are present, biopsies will be taken both from an injected tumor and a non-injected tumor and a comparison will be done between them. We will generate a patient-specific profile of tumor microenvironment. We will identify the cell types that are present in each patient at onset of treatment and how cellular composition changes in response to treatment. By immunostaining, flow cytometry or RNA sequencing using computational approaches we will cluster the cells from each sample by their expression profile to distinct groups representing specific cell types (e.g. tumor cells, lymphocytes, CD45+, squamous epithelium). Similarly, we will identify various immune cells such as but not limited at, CD8+ and CD4+, effector T cells, T<sub>reg</sub> and others immune subtypes and correlate with microbiome composition. Using this data, we will try to find correlates between different tumor-immune microenvironment components and clinical outcome. In addition, we will survey levels of PD-1, PD-L1/2, CD28 and other known marker of checkpoint inhibitor response.

We will correlate the responses to the oncolytic virus with the presence/absence of the stromal changes using a Fisher exact test.

# B. Longitudinal profiling of patients before and after immunotherapy + OBP-301 + SBRT to identify possible biomarkers for response and mechanism of resistance

We will do longitudinal profiling of patients before and after immunotherapy + OBP-301 to identify possible biomarkers for response and mechanism of resistance.

We plan to investigate different biomarkers i.e. circulating tumor DNA (ctDNA) and tumor and plasma exosomes.

**B1**. The Cancer Genome Atlas demonstrated that specific genes and pathways are commonly altered in head and neck cancer, namely *TP53*, *NOTCH1*, *PIK3CA*, among other genes<sup>69</sup>. Also, predictable genetic alterations underlie HPV positive HNSCCs, such as the presence of HPV-16 viral DNA, p16<sup>INK4A</sup> overexpression. Researchers have found HPV DNA present in blood<sup>70</sup>, offering the possibility of a simple blood draw or saliva swab to detect cancer.

We will investigate the utility of using ctDNA and exosomes both in HPV positive and HPV negative tumors to monitor response after immunotherapy + OBP-301 + SBRT.

We will correlate the responses to the oncolytic virus with the presence/absence of the ctDNA changes using a Fisher exact test.

**B2**. Another potentially interesting biomarkers are exosomes. The cargo of plasma exosomes from head and neck patients may contain valuable biomarkers with predictive value for head and neck cancer progression and response to therapies. Blood and tissue will be obtained from patients. Tissue will be obtained from prior surgeries. Tissue will be examined for extracellular matrix composition and cellular infiltrate using immunofluorescence (IF, classical or Hyperion mass cytometry based), immuno-histochemistry (IHC) or flow cytometry. Blood will be placed into EDTA coated tubes and centrifuged at 500 x g for 10 minutes at 4°C, followed by a second centrifugation step at 3000 x g for 20 minutes at 4°C and plasma will be stored at -80°C until the time of analysis. Tissues will be embedded in paraffin as well as O.C.T. and frozen.

At the time of analysis, which will be performed in the lab of Dr. David Lyden at Weill Cornell Medical College/Cornell University, exosomes will be isolated from plasma, media from tumor biopsy tissue cultures by serially ultracentrifugation. Exosome size and number will be quantified using nanoparticle tracking analysis (Nanosight®, Malvern), and exosome cargo will be characterized using genomic and proteomic approaches (DNA/RNA sequencing, real-time PCR and mass spectrometry, Western blot or Elisa).

We will correlate the responses to the oncolytic virus with exosome number, size and cargo changes using a Fisher exact test.

We will summarize the results from all patient data to assess what are the consistent changes observed in biomarkers in response to immunotherapy and we will investigate how these biomarkers are related to response to treatment.

# C. To examine and characterize the immune infiltrate by multi-parameter flow-cytometry

In this application, innovative multi-parameter flow cytometry will be utilized that will provide single-cell high resolution of immune cell suppression or activation. Investigators in Weill Cornell have developed technologies to cryopreserve viable immune cells from primary human tissues and tumor biopsies or resections for side-by-side analyses of immune cells from multiple patients, thus reducing sample variation and allowing direct single-cell comparisons of cytokine production. This approach will be utilized to characterize tumor immune cell infiltrates at baseline, following the induction of combination therapy and at the time of resection. This will be one of the first longitudinal analyses of tumor immune cell infiltrates by multi-parameter flow cytometry following immunotherapy. To examine and characterize the phenotype of immune infiltrates.

We will correlate the responses to the oncolytic virus with the presence/absence of immune infiltrates changes using a Fisher exact test.

# D. To investigate the presence of circulating tumor cells before, after treatment and at recurrence/progression in the blood using TelomeScan Telomescan.

TelomeScan (OBP-401) a new telomerase-based liquid biopsy biomarker, will be used to detect the presence of circulating tumor cells in the blood. This technique allows the specific staining of circulating blood will be drawn before beginning of treatment, after completion of SBRT and at recurrence/progression.

The blood sample processing for sequential monitoring of circulating tumor cells (CTCs)analysis using TelomeScan is described in the Standard Operation Procedure is included as appendix A.

| Specimen type | Timepoint |
|-------------------|----------------------------------|
| ACD tube x1 8.5ml | Screening |
| 0.31111 | Day 1 |
| | Day 8 |
| | Day 18 |
| | Day 22 |
| | Day 94 |
| | Upon progression or end of study |

We will correlate the responses to the oncolytic virus with the presence/absence of CTCs in the peripheral blood using a Fisher exact test.

#### 10.7 Safety Analyses

#### 10.7.1 Safety Endpoints

The primary safety endpoint is to examine the safety of multiple OBP-301 intratumoral injections in combination with pembrolizumab in advanced esophagogastric cancer.

#### 10.7.2 Summary of Adverse Events

All adverse events, will be recorded for each patient. Adverse events will be tabulated for all patients by: first occurrence of each adverse event, maximum severity, and relationship to treatment. Treatment-related AEs and serious AEs will be tabulated separately, by first occurrence, maximum severity, and strongest relationship to treatment. A listing of all AEs

will also be included, per patient, including onset/resolution date, severity, relationship to study treatment, and action regarding IP. A listing of all discontinuations, injection delays, and deaths due to adverse events in the study will be included.

#### 10.7.3 Summary of Laboratory Assessments

Summary statistics will be presented for all blood chemistry, hematology, coagulation, and urinalysis results by study visit, where data are collected.

In addition, all laboratory values will be flagged as low (L1, L2, L3, or L4), high (H1, H2, H3, or H4) or normal (N) based on the investigational site laboratory normal range and/or the NCI toxicity criteria. Shifts in assessments from baseline to all post-baseline visits will be presented (shift tables).

#### 10.7.4 Summary of Special Laboratory Assessments

Summary statistics and shift tables will be presented for all special laboratories results including cytokines, and immune cell phenotypes by study visit, where data are collected.

#### 10.7.5 Summary of Vital Signs

Summary statistics will be presented for all vital signs including temperature, blood pressure (systolic and diastolic), pulse, respiration rate, and body weight by study visit, where data are collected. Graphs of vital signs at each visit may also be provided.

#### 10.7.6 Summary of Physical Examinations

The physical examination results will be evaluated by shift tables that compare baseline examination results to other study visit results in each exam. Frequency counts and percentages will be displayed. All abnormal results will be provided in a listing with a description of the abnormality.

#### **10.7.7** Summary of ECG Measurements

The results of the ECG will be evaluated by transition tables that compare Screening exam results to Final Visit results. Frequency counts and percentages will be displayed. All abnormal results will be provided in a listing with a description of the abnormality.

#### 10.7.8 Concomitant Medications

Concomitant medications will be tabulated for all patients by: the first occurrence of medication classes, the first occurrence of concomitant medications, and all concomitant medications. A listing of all concomitant medications will also be provided.

# 10.7.9 Adverse Event Stopping Rule

The stopping rule specified below is based on the knowledge available at study development. We note that the Adverse Event Stopping Rule may be adjusted in the event of either (1) the study re-opening to accrual or (2) at any time during the conduct of the trial and in consideration of newly acquired information regarding the adverse event profile of the treatment(s) under investigation. The study team may choose to suspend accrual because of unexpected adverse event profiles that have not crossed the specified rule below.

Accrual will be temporarily suspended to the study to allow for a full review of data according to the following AE stopping rule:

(1)If, at any time, more than 3 of the first 12 patients enrolled (or  $\geq$  33% of all patients enrolled after 12 patients) have experience at least one grade 3 or worse immune related adverse event or adverse event related (possibly, probably, or definitely) to OBP-301 injection.

Immune related adverse events for the purposes of this adverse event stopping rule, will include diarrhea/colitis, pneumonitis, renal failure/nephritis, or increased LFTS (bilirubin, AST, ALT). Rash, joint aches, fatigue, thyroid abnormalities, or other immune related events that are not life threatening will not be included for the purposes of this Adverse Event Stopping Rule.

- (2) If grade 5 (death) event at least possibly, probably or definitely related to OBP-301 injection, the study will be halted.
- (3) If 3 or more grade 4 adverse events that are possibly, probably, or definitely attributed to OBP-301 occur, that do not resolve back to grade 1 within 30 days, the study will be halted.

#### 10.7.10 Adverse Event Dose De-escalation

If, after the first injection of OBP-301, 3 of the first 12 patients enrolled have experienced at least one grade 3 or worse immune related adverse event or adverse event related (possibly, probably, or definitely) to OBP-301 injection i.e. rash, joint aches, fatigue, thyroid abnormalities, or other immune related events that are not life threatening the concentration of OBP-301 will be reduced from  $1 \times 10^{12}$  VP/mL to  $1 \times 10^{11}$  VP/mL. Further de-escalation will be considered (i.e decrease of the number of OBP-301 injections by 25%) if more patients develop after the first injection at least one grade 3 or worse immune related adverse event or adverse event related (possibly, probably, or definitely) to OBP-301 injection i.e. rash, joint aches, fatigue, thyroid abnormalities, or other immune related events.

If needed, OBP-301 dose level will be DE-ESCALATED to  $1 \times 10^{11}$  viral particles (vp)/mL (up to 4 mL of OBP-301 should be injected based on the tumor volume)) per intra-tumoral injection.

The following **dilution instructions** will be used:

#### 10.7.11 OBP-301 10x Dilution Procedure:

- 1. Preparation Step: Use injection syringe to suck the 1 ml from 1x10^12 vp/mL vial. and use diluted solution syringe to suck the 9 mL D5W (Dextrose 5% in Water).
- 2. Dilution Step: Slowly push 1 mL OBP-301 to Diluted solution syringe, and vertically mix in gentle motion for 20 times (The concentration of diluted solution syringe would be 1 x 10^11 vp/mL).



Injection syringe T shape stopcock Or luer lock connector Diluted solution (D5W) syringe

1 mL 9 mL

# 10.8 Determination of Sample Size

#### Phase II study:

#### **Statistical Considerations:**

The primary endpoint for this study will be the objective response rate (CR + PR). Sample size recommendations for the phase II design are determined according to Simon's two-stage design (Simon R, 1989). We project an objective response proportion of 61%, below which the response will be unacceptable, and an objective response proportion of 78%, above which the regimen will be considered worthy of further exploration. The null hypothesis that the objective response proportion is less than or equal to 61% will be tested against the alternative hypothesis that the response proportion is greater than or equal to 78%.

The sample size computations were performed assuming 10% level of significance and 80% power. In the first stage, 12 patients will enter the study. If 7 or fewer respond, the study will be terminated early and declared to have a negative result. If 8 or more patients respond, enrollment will be extended to 36 patients. At Stage 2, the treatment will be declared effective and worthy of further testing if 26 or more patients respond among the 36 patients entered. This two-stage design yields a  $\geq 0.80$  probability of a positive result if the true percentage of overall responders is  $\geq 78\%$ . It yields a  $\geq 0.90$  probability of a negative result if the true percentage of overall responders is  $\leq 61\%$ . A 95% confidence interval constructed around the expected objective response proportion of 78% can be estimated to be within  $\pm$  16.0% of the observed response proportion.

Assuming 10% are unevaluable/ineligible, we anticipate that a total of 14 patients will be enrolled in the first stage, 40 in both the first and second stage if the study proceeds to the second stage.

**Table 1.** Numbers of observed responders required to accept or reject H0 at each stage. Under this design, H0 will not be rejected at Stage 1.

| | N | Accept H <sub>0</sub> | Reject H <sub>0</sub> |
|---------|----|-----------------------|-----------------------|
| Stage 1 | 12 | ≤ 7 | |
| Stage 2 | 36 | ≤ 25 | >26 |

Analysis Plan for Endpoints:

## **Primary Endpoint:**

The primary endpoint of objective response rate (CR + PR) will be estimated and a 95% confidence interval will be estimated via binomial proportions.

### **Secondary Clinical Endpoints:**

With adequate follow-up time, secondary endpoints of progression-free survival (PFS) and overall survival (OS) will be assessed by Kaplan-Meier survival analysis and 95% confidence intervals will be calculated using Greenwood's formulae. PFS will be defined as the time from first treatment day until objective or symptomatic progression or death. OS will be defined as the time from first treatment day until death.

The frequency of subjects experiencing toxicities in each treatment arm will be tabulated. Toxicities will be assessed and graded according to CTCAE v. 5.0 terminology. Exact 95% confidence intervals around the toxicity proportions will be calculated to assess the precision of the obtained estimates.

All analyses will be performed in SAS Version 9.4 (SAS Institute, Inc., Cary, North Carolina) and Stata Version 15.0 (Stata Corporation, College Station, Texas). For Reference of the Phase 2 design see 41.

# **Analysis Plan for Endpoints:**

### Primary Endpoint:

The primary end point is the objective response rate (ORR) according to RECIST v. 1.1 of multiple OBP-301 intratumoral injections in combination with pembrolizumab in recurrent locally advanced head and neck cancer. The frequency of subjects experiencing toxicities will be tabulated. Toxicities will be assessed and graded according to CTCAE v 5.0 terminology.

#### Secondary endpoints:

Secondary endpoints include the OS proportion at 1 year, the Kaplan-Meier progression free survival (PFS) and the toxicity profile of this three treatments combination. Median OS, including survival curves, will be estimated using Kaplan-Meier methodology. Greenwood's formula will be used to calculate 95% confidence intervals for the Kaplan-Meier estimates.

All analyses will be performed in SAS Version 9.4 (SAS Institute, Inc., Cary, North Carolina) and Stata Version 15.0 (Stata Corporation, College Station, Texas).

#### 11 REGULATORY REQUIREMENTS

#### 11.1 Regulatory Approvals

Once protocol amendments or consent form modifications are implemented at the lead site, Weill Cornell Medicine, updated documents will be provided to participating sites. Weill Cornell Medicine must approve all consent form changes prior to local IRB submission.

Relevant study documentation will be submitted to the regulatory authorities of the participating countries, according to local/national requirements, for review and approval before the beginning of the study. On completion of the study, the regulatory authorities will be notified that the study has ended.

As required by local regulations, the Investigator will ensure all legal aspects are covered, and approval of the appropriate regulatory bodies obtained, before study initiation.

## 11.2 Institutional Review Board/Ethics Committee Approval

Before initiation of the study at each study center, the protocol, the ICF, other written material given to the patients, and any other relevant study documentation will be submitted to the appropriate Ethics Committee. Written approval of the study and all relevant study information must be obtained before the study center can be initiated or the IP is released to the Investigator. Any necessary extensions or renewals of IEC/IRB approval must be obtained for changes to the study, such as amendments to the protocol, the ICF, or other study documentation. The written approval of the IEC/IRB together with the approved ICF must be filed in the study files.

The Investigator will report promptly to the IEC/IRB any new information that may adversely affect the safety of the patients or the conduct of the study. The Investigator will submit written summaries of the study status to the IEC/IRB as required. On completion of the study, the IEC/IRB will be notified that the study has ended.

Neither the Investigator nor Oncolys BioPharma Inc. will modify or alter this protocol without the agreement of the other. All agreed protocol amendments will be clearly recorded on a protocol amendment form and will be signed and dated by the original protocol approving signatories. All protocol amendments will be submitted to the relevant institutional IEC/IRB for approval before implementation, as required by local regulations. The only exception will be when the amendment is necessary to eliminate an immediate hazard to the trial participants. In this case, the necessary action will be taken first, with the relevant protocol amendment following shortly thereafter.

#### 11.3 Ethical Conduct of the Study

The Investigators and all parties involved should conduct this study in adherence to the ethical principles based on the Declaration of Helsinki, GCP, ICH guidelines and the applicable national and local laws and regulatory requirements.

This study will be conducted under a protocol reviewed and approved by the applicable ethics committees and investigations will be undertaken by scientifically and medically qualified persons, where the benefits of the study are in proportion to the risks.

# 11.4 Participant Informed Consent

The Investigator is responsible for ensuring that no subject undergoes any study-related examination or activity before that subject has given written informed consent to participate in the study.

It is the Investigator's responsibility to ensure that each participant gives informed consent to participate in the study. The Investigator will explain the nature of the study, its purpose, procedures, expected duration, and the potential benefits, risks and inconveniences in participation. In addition, a participant information sheet/consent form containing relevant information will be prepared by Oncolys BioPharma Inc. in conjunction with the investigational site and will be provided to all participants.

Participants must be informed that their participation is voluntary and that they have the right to withdraw from the study at any time without prejudice.

The participants will be informed of their rights to privacy but will be made aware that the study data will be submitted to Oncolys BioPharma Inc. and possibly to drug regulatory authorities for review and evaluation. They will be informed also that the study monitor may inspect their medical records to verify the accuracy and completeness of the study records and results.

The ICF will contain a separate section that addresses the use of remaining blood and tissue samples for future research. Participants will be informed that they are free to refuse to these additional tests being carried out and may request at any time for the samples to be destroyed.

The participants will be given an opportunity to ask questions and allowed sufficient time to decide whether they wish to participate. If the participant decides to participate in the study, they will voluntarily sign the written ICF.

The acquisition of informed consent should be documented in the participant's medical records, and should meet the requirements of GCP. The ICF will be signed and personally dated by the participant and by the person who conducted the informed consent discussion (not necessarily an Investigator). The original signed ICF will be retained in accordance with institutional policy, and a copy of the signed consent form will be provided to the participant or legal representative. The date that informed consent was signed will be recorded on the eCRF.

If new information becomes available that may be relevant to the patient's willingness to continue participation in the study, the ICF will be updated and approved by the IEC(s)/IRB(s) (and regulatory authorities, if required). The study participants will be informed about this new information and reconsent will be obtained.

Participants who are rescreened are required to sign a new ICF.

#### 11.5 Compliance with Trial Registration and Results Posting Requirements

Under the terms of the Food and Drug Administration Modernization Act (FDAMA) and the Food and Drug Administration Amendments Act (FDAAA), the Sponsor-Investigator of the trial is solely responsible for determining whether the trial and its results are subject to the requirements for submission to http://www.clinicaltrials.gov. Information posted will allow subjects to identify potentially appropriate trials for their disease conditions and pursue

participation by calling a central contact number for further information on appropriate trial locations and trial site contact information.

#### 12 DATA AND SAFETY MONITORING PLAN (DSMP)

**12.1** The study will be reviewed by the Weill Cornell Medical College Data and Safety Monitoring Board (DSMB) as an independent means of data and safety monitoring. Enrollment information, adverse event and safety information, protocol changes, and other interim data will be evaluated by the DSMB. After each evaluation, the Board will provide the principal investigator with recommendations for protocol modification, continuation, or termination.

DSMB reports will be made to the DSMB every 6 months.

### 12.2 The radiotherapy safety monitoring committee (RSMC)

In order to avoid radiation toxicities, an independent safety monitoring committee formed by several radiation oncologists with expertise in the SBRT techniques and not involved in the study will review all radiotherapy treatment plans.

#### 13 ADMINISTRATIVE PROCEDURES

#### 13.1 Financing, Liability/Indemnity/Insurance

Investigators are required to follow financial disclosure policies at their respective institutions. Any investigator with a conflict of interest with this study must report the conflict to the Sponsor-investigator.

The study contract will govern all provisions relating to liability, indemnity and insurance.

#### 13.2 Recording of Data and Retention of Records

Essential documents are those documents that individually and collectively permit evaluation of the study and quality of the data produced. After completion of the study (end of study defined as the date of the last follow-up contact at Week 48 with the last patient), all documents and data relating to the study will be kept in an orderly manner by the Investigator in a secure study file. Essential documents should be retained for 2 years after the final marketing approval in an ICH region or for at least 2 years since the discontinuation of clinical development of the IP. In addition, all patient medical records and other source documentation will be kept for the maximum time permitted by the hospital, institution, or medical practice.

# **13.2.1 REDCap**

REDCap (Research Electronic Data Capture) is a free data management software system that is fully supported by the Weill Cornell Medical Center CTSC. It is a tool for the creation of customized, secure data management systems that include Web-based data-entry forms, reporting tools, and a full array of security features including user and group based privileges, authentication using institution LDAP system, with a full audit trail of data manipulation and export procedures. REDCap is maintained on CTSC-owned servers that are backed up nightly and support encrypted (SSL-based) connections. Nationally, the software is developed,

enhanced and supported through a multi-institutional consortium led by the Vanderbilt University CTSA.

#### 13.3 Retention of Records

Essential documents are those documents that individually and collectively permit evaluation of the study and quality of the data produced. After completion of the study (end of study defined as the date of the last follow-up contact at Week 48 with the last patient), all documents and data relating to the study will be kept in an orderly manner by the Investigator in a secure study file. Essential documents should be retained for 2 years after the final marketing approval in an ICH region or for at least 2 years since the discontinuation of clinical development of the IP. In addition, all patient medical records and other source documentation will be kept for the maximum time permitted by the hospital, institution, or medical practice.

#### 13.4 Disclosure and Data Confidentiality

The Investigator must ensure that the participant's anonymity is maintained. Participants should only be identified by their initials and a participant identification number on the eCRFs and other source documents. Other study-related documents (e.g., signed ICFs) should be kept in strict confidence by the Investigator.

Data is captured using database REDCap. Participants will be informed that data will be held on file by Oncolys BioPharma Inc. and that these data may be viewed by staff including the study monitor and by external auditors on behalf of Oncolys BioPharma Inc. and appropriate regulatory authorities. Participants will also be informed that a study report will be prepared and may be submitted to regulatory authorities and for publication. However, participants will be identified in such reports only by study identification number, gender, and age. All participant data will be held in strict confidence.

Auditors, the IEC(s)/IRB(s) approving this research, and the US FDA, as well as that of any other applicable agency(ies), will be granted direct access to the study patients' original medical records for verification of clinical study procedures and/or data, without violating the confidentiality of the patients to the extent permitted by the law and regulations. In any presentations of the results of this study or in publications, the patients' identity will remain confidential.

All personal data collected and processed for the purposes of this study should be managed by the Investigator and his/her staff with adequate precautions to ensure confidentiality of those data, and in accordance with the HIPAA<sup>64</sup>, applicable to national and/or local laws and regulations on personal data protection.

#### 13.5 Publication of Results

Study results will be reported at appropriate international congresses and meetings as data are available, and the final study will be reported in a peer-reviewed oncology journal.

#### 14 CLINICAL STUDY REPORT

We will provide the clinical study report to Oncolys Biopharma within 1 year of study completion.

# 15 APPENDICES

# 15.1 ECOG performance status

| Performance<br>Status | Definition |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without restriction. |
| 1 | Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work. |
| 2 | Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours. |
| 3 | Capable of limited self-care, confined to bed or chair more than 50% of waking hours. |
| 4 | Completely disabled; cannot carry on any self-care; totally confined to bed or chair. |

# 15.2 Comparison of RECIST 1.1 and iRECIST

| | RECIST 1.1 | iRECIST |
|---|---|---|
| Definitions of | Measurable lesions are ≥10 | No change from RECIST 1.1; |
| measurable and | mm in diameter (≥15 mm for | however, new lesions are assessed |
| non-measurable | nodal lesions); maximum of | as per RECIST 1.1 but are recorded |
| disease; numbers | five lesions (two per organ); | separately on the case report form |
| and site of target | all other disease is considered | (but not included in the sum of |
| disease | non-target (must be ≥10 mm | lesions for target lesions identified at |
| | in short axis for nodal | baseline) |
| | disease) | |
| Complete | Cannot have met criteria for | Can have had iUPD (one or more |
| response, partial | progression before complete | instances), but not iCPD, before |
| response, or stable | response, partial response, or | iCR, iPR, or iSD |
| disease | stable disease | |
| Confirmation of | Only required for non- | As per RECIST 1.1 |
| complete response | randomized trials | |
| or partial response | | |
| Confirmation of | Not required | As per RECIST 1.1 |
| stable disease | | |
| New lesions | Result in progression; | Results in iUPD but iCPD is only |
| | recorded but not measured | assigned on the basis of this |
| | | category if at next assessment |
| | | additional new lesions appear or an |

| | | increase in size of new lesions is seen (≥5 mm for sum of new lesion target or any increase in new lesion non-target); the appearance of new lesions when none have previously been recorded, can also confirm iCPD |
|---|---|---|
| Independent<br>blinded review and<br>central collection<br>of scans | Recommended in some circumstances—i.e., in some trials with progression-based endpoints planned for marketing approval | Collection of scans (but not independent review) recommended for all trials |
| Confirmation of progression | Not required (unless equivocal) | Required |
| Consideration of clinical status | Not included in assessment | Clinical stability is considered when deciding whether treatment is continued after iUPD |

<sup>&</sup>quot;i" indicates immune responses assigned using iRECIST. RECIST=Response Evaluation Criteria in Solid Tumours. iUPD=unconfirmed progression. iCPD=confirmed progression. iCR=complete response. iPR=partial response. iSD=stable disease.

# 15.3 Appendix

See attached Informed Consent and Clinical Trials Monitoring Plan including the SBRT Safety form.

#### 14. REFERENCES:

- 1. Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012;12(4):252-264.
- 2. Brahmer JR, Tykodi SS, Chow LQ, et al. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012;366(26):2455-2465.
- 3. Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, al. e. Safety, activity, and immunecorrelates of anti-PD-1 antibody in cancer. N Engl J Med. 2012;366(26):2443-2454.
- 4. Robert C, Long GV, Brady B, Dutriaux C, Maio M, al. e. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med. 2015;372(4):320-330.
- 5. Robert C, Schachter J, Long GV, et al. pembrolizumab versus ipilumumab in advanced melanoma. N Engl J Med. 2015;372(26):2521-2532.
- 6. Brahmer J, Reckamp KL, Bass P, Crino L, Eberhardt WE, al. e. Nivolumab versus docetaxel in advanced squamous-cell non-small-cell lung cancer. N Engl J Med. 2015;373(2):123-135.

7. Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, al. e. Nivolumab versus docetaxel in advanced nonsquamous non-small-cell lung cancer. N Engl J Med. 2015;373(17):1627-1639.

- 8. Garon EB, Rizvi NA, Hui R, Leighl N, Balmonoukian AS, al. e. pembrolizumab for the treatmnt of non-small cell lung cancer. N Engl J Med. 2015;372(21):2018-2028.
- 9. Reck M, Rodriquez-Abreu D, Robinson AG, et al. pembrolizumab versus chemothreapy for PD-L1 positive non-small cell lung cancer. N Engl J Med. 2016;375(19):1823-1833.
- 10. Motzer RJ, Escudier B, McDermott DF, et al. Nivolumab versus everolimus in advanced renal-cell carcinoma. N Engl J Med. 2015;373(19):1803-1813.
- 13. Chow LQM, et al. Antitumor Activity of pembrolizumab in Biomarker-Unselected Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma: Results From the Phase Ib KEYNOTE-012 Expansion Cohort. J Clin Oncol 34 (32) (November 2016) 3838-3845.
- 14. Bauml J, et al. pembrolizumab for Platinum- and Cetuximab-Refractory Head and Neck Cancer: Results From a Single-Arm, Phase II Study. J Clin Oncol. 2017 May 10; 35(14): 1542–1549.
- 15. Ferris, RL et al. Nivolumab for Recurrent Squamous-Cell Carcinoma of the Head and Neck N Engl J Med 2016; 375:1856-1867.
- 16. Ferris RL, et al. Nivolumab vs investigator's choice in recurrent or metastatic squamous cell carcinoma of the head and neck: 2-year long-term survival update of CheckMate 141 with analyses by tumor PD-L1 expression. Oral Oncology 2018; 81:45-51.
- 17. R. Bahleda, F.S. Braiteh, A.S. Balmanoukian, I. Braña, F. S. Hodi, L. Garbo, B. Liu, L. Molinero, C. O'Hear, X. Shen, M. Fasso, A.D. Colevas Long-Term Safety and Clinical Outcomes of pembrolizumab in Head and Neck Cancer: Phase Ia Trial Results Annals of Oncology (2017) 28 (suppl\_5): v372-v394.
- 18. D. Zandberg, A. Algazi, A. Jimeno<sup>3</sup>, J.S. Good, J. Fayette, N. Bouganim, N. Ready, P.M. Clement, T. Goswmi, A. Jarkowski, J.M. Armstrong, K. Asubonteng, G. Melillo, R. Mesía 1042O Durvalumab for recurrent/metastatic (R/M) head and neck squamous cell carcinoma (HNSCC): preliminary results from a single-arm, phase 2 study Annals of Oncology (2017) 28 (suppl\_5): v372-v394.
- 19. Kaufman HL, Kohlhapp FJ, Zloza A. Oncolytic viruses: a new class of immunotherapy drugs. Nat ReDrug Discov. 2015; 14 (9):642-662.
- 20. Kawashima T, Kagawa S, Kobayashi N, al. e. Telomerase-specific replication-selective virotherapy in human cancer. Clin Cancer Res. 2004;10:285-292.
- 21. Umeoka T, Kawashima T, Kagawa S, al. e. Visualization of intrathoracically disseminated solid tumors in mice withoptical imaging by telomerase-specific amplification of a transferred gene fluorescent protein gene. Cancer Res. 2004;64(6259-65.).

- 22. Taki M, Kagawa S, Nishizaki M, al. e. Enhanced oncolysis by a tropism-modified telomerase-specific replication-selective adenoviral agent OBP-405 (Telomyelysin-RGD). Oncogene. 2005;24:3130-3140.
- 23. Hashimoto Y, Watanabe Y, Shirakiya Y, al. e. Establishment of biological and pharmacokinetic assays of telomerase-specific replication-selective adenovirus. Cancer Sci. 2008;99(385-90.).
- 24. Nemunaitis JJ, Tong AW, Nemunaitis M, Senzer N, Phadke AP, al. e. A phase I study of telomerase-specific replication competent oncolytic adenovirus (OBP-301) for various solid tumors. Mol Ther. 2010;18(2):429-434.
- 25. Sharma P, Allison JP. The future of immune checkpoint therapy. Science. 2015;348(6230):56-61.
- 26. Hellmann MD, Friedman CF, Wolchok JD. Combinatorial cancer immunotherapies. Adv Immunol. 2016;130:251-277.
- 27. Zou W, Wolchok JD, Chen L. PD-L1 (B7-H1) and PD-1 pathway blockade for cancer therapy: Mechanisms, response biomarkers, and combinations. Sci Transl Med. 2016;8(328):328rv324.
- 28. Chen L, Han X. Anti-PD-1/PD-L1 therapy of human cancer: past, present, and future. J Clin Invest. 2015;125(9):3384-3391.
- 29. Minn AJ, Wherry EJ. Combination cancer therapies with immune checkpoint blockade: convergence on interferon signaling. Cell. 2016;165(2):272-275.
- 30. Hepworth MR, Fung TC, Masur SH, Kelsen JR, McConnell FM, al. e. Immune tolerance. Group 3 innate lymphoid cells mediate intestinal selection of commensal bacteria-specific CD4+ T cells. Science. 2015;348(6238):1031-1035.
- 31. Withers DR, Hepworth MR, Wang X, Mackley EC, Halford EE, al. e. Transient inhibition of ROR-vt therapeutically limits intestinal inflammation by reducing TH17 cells and preserving group 3 innate lymphoid cells. Nat Med. 2016;22(3):319-323.
- 32. Comet B, Kramar A, Faivre-Pierret M, et al. Salvage stereotactic reirradiation with or without cetuximab for locally recurrent head-and-neck cancer: a feasibility study. Int J Radiat Oncol Biol Phys. 2012;84(1):203-209.
- 33. Lartigau EF, Tresch E, Thariat J, et al. Multi institutional phase II study of concomitant stereotactic reirradiation and cetuximab for recurrent head and neck cancer. Radiother Oncol. 2013;109 (2):281-285.
- 34. Kodani N, Yamazaki H, Tsubokura T, et al. Stereotactic body radiation therapy for head and neck tumor: disease control and morbidity outcomes. J Radiat Res 2011;52:24–31.
- 35. Roh KW, Jang JS, Kim MS, et al. Fractionated stereotactic radiotherapy as reirradiation for locally recurrent head and neck cancer. Int J Radiat Oncol Biol Phys. 2009;74(5):1348-1355.
- 36. Zafereo ME, Hanasono MM, Rosenthal DI et al. The role of salvage surgery in patients with recurrent squamous cell carcinoma of the oropharynx. Cancer 115(24), 5723–5733 (2009).

- 37. Vermorken JB, Mesia R, Rivera F et al. Platinum-based chemotherapy plus cetuximab in head and neck cancer. N. Engl. J. Med. 359(11), 1116–1127 (2008).
- 38. Vermorken JB, Remenar E, Hitt R, Kawecki A, Rottey S, Knierim L, et al. Platinum-based chemotherapy (CT) plus cetuximab in recurrent or metastatic squamous cell carcinoma of the head and neck cancer (R/M-SCCHN): 5-year follow-up data for the extreme trial. J Clin Oncol. 2014;32(suppl):abstr 6021.
- 39. Peiffert D, Pernot M, Malissard L et al. Salvage irradiation by brachytherapy of velotonsillar squamous cell carcinoma in a previously irradiated field: results in 73 cases. Int. J. Radiat. Oncol. Biol. Phys. 29(4), 681–686 (1994).
- 40. Simon J Dovedi, Eleanor J Cheadle, Amy Popple, et al. Fractionated radiation therapy stimulates anti-tumor immunity mediated by both resident and infiltrating polyclonal T-cell populations when combined with PD1 blockade. Clin Cancer Research 2017. 23. 5514-5523.
- 41. Simon R (1989): Optimal Two-Stage Designs for Phase II Clinical Trials, Controlled Clinical Trials, 10:1-10.
- 42. Krcik EM. Radiation Therapy Plus Anti-Programmed Death Ligand 1 Immunotherapy: A Review on Overall Survival. Radiol Technol. 2016 Sep;88(1):123-8.
- 43. Kanaya N et. Al. Abstract 2744 AACR 2018.
- 44. Kojima et. Al. Abstract # 7607 AACR 2019.
- 45. Tanabe S, et al. J Clin Oncol. 2019;37(4)\_suppl:130.
- 46. Harrington, K. J. et al. Safety and preliminary efficacy of talimogene laherparepvec (T-VEC) in combination (combo) with pembrolizumab (pembro) in patients (pts) with recurrent or metastatic squamous cell carcinoma of the head and neck (R/M HNSCC): a multicenter, phase 1b study (MASTERKEY-232) [abstract]. J. Clin. Oncol. 2018. 36 (Suppl. 15), 6036.
- 47. Harrington K, et al. Optimizing oncolytic virotherapy in cancer treatment. Nat Rev Drug Discov. 2019 Sep; 18(9):689-706.
- 48. Koujima T, Tazawa H, Ieda T, Araki H, Fushimi T, Shoji R, Kuroda S, Kikuchi S, Yoshida R, Umeda Y, Teraishi F, Urata Y, Mizuguchi H, Fujiwara T, Oncolytic Virus-Mediated Targeting of the ERK Signaling Pathway Inhibits Invasive Propensity in Human Pancreatic Cancer, *Molecular Therapy: Oncolytics* (2020), doi: https://doi.org/10.1016/j.omto.2020.03.016.
- 49. Andtbacka, R.H., et al., Talimogene Laherparepvec Improves Durable Response Rate in Patients With Advanced Melanoma. J Clin Oncol, 2015. 33(25): 2780-8.
- 50. Goodin, T., FDA approves first-of-its-kind product for the treatment of melanoma, in FDA News Release. 2015 (page 1).
- 51. Benstetter, M., First oncolytic immunotherapy medicine recommended for approval, in European Medicines Agency Press Release. 2015 (page 1).

52. Hawkins, L.K., et al., Gene delivery from the E3 region of replicating human adenovirus: evaluation of the 6.7 K/gp19 K region. Gene Ther, 2001. 8(15): 1123-31.

- 53. Shay, J.W. and S. Bacchetti, A survey of telomerase activity in human cancer. Eur J Cancer, 1997. 33(5): 787-91.
- 54. Shay, J.W., et al., Telomerase and cancer. Hum Mol Genet, 2001. 10(7): p. 677-85.
- 55. Kamradt, J., et al., Telomerase activity and telomerase subunit gene expression levels are not related in prostate cancer: a real-time quantification and in situ hybridization study. Lab Invest, 2003. 83(5): 623-33.
- 60. OBP-301 OBP-301. Investigator's Brochure, version 8.0, O.B. Inc, Editor. 2017.
- 61. Sub-analysis Report of OBP-301 Phase I study in patients with Melanoma, Study Number: 0301-1-0002. Implementation period: 2016/1/12-2016/1/15. 2016, Oncolys BioPharma Inc.
- 62. Song, X., et al., Overall survival in patients with metastatic melanoma. Curr Med Res Opin, 2015. 31(5): 987-91.
- 63. Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 U.D.o.H.a.H.S.N.I.o.H.N.C. Institute, Editor. 2010.
- 64. Services, U.D.o.H.a.u., The Health Insurance Portability and Accountability Act (HIPAA) of 1996 (P.L. 104-191) [HIPAA 1996].
- 65. Lang, FF et al. Phase I Study of DNX-2401 (Delta-24-RGD) Oncolytic Adenovirus: Replication and Immunotherapeutic Effects in Recurrent Malignant Glioma. J Clin Oncol. 2018. 36:1419-1427.
- 66. Fujiwara, T. Multidisciplinary oncolytic virotherapy for gastrointestinal cancer. Ann Gastroenterol Surg. 2019;3:396–404.
- 67. Burtess, B et al. Pembrolizumab alone or with chemotherapy versus cetuximab with chemotherapy for recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-048): a randomised, open-label, phase 3 study. Lancet. 2019, 394(10212):1915-1928.
- 68. Seki, T et al. Fiber shaft extension in combination with HI loop ligands augments infectivity for CAR-negative tumor targets but does not enhance hepatotropism in vivo. Gene Therapy. 2002; 9: 1101–1108.
- 69. Cancer Genome Atlas N. Comprehensive genomic characterization of head and neck squamous cell carcinomas. 2015. Nature 517 (7536):576–582.
- 70. Jensen KK, Grønhøj C, Jensen DH, von Buchwald C. Circulating human papillomavirus DNA as a surveillance tool in head and neck squamous cell carcinoma: A systematic review and meta-analysis. Clin Otolaryngol. 2018. 43(5):1242-1249.

71. Baliga, S, Kabarriti, R, Ohri, N, et al. Stereotactic body radiotherapy for recurrent head and neck cancer: A critical review. Head Neck. 39(3):595-601.